

#### STATISTICAL ANALYSIS PLAN

**Study Title:** A Phase 3b, Randomized, Open-Label Study to Evaluate the

Safety and Efficacy of Switching from Regimens Consisting of Abacavir/Lamivudine (ABC/3TC) plus a Third Antiretroviral Agent to the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Fixed-Dose Combination (FDC) in Virologically-Suppressed HIV-1 Infected Adult Subjects

Name of Test Drug: E/C/F/TAF FDC

Study Number: GS-US-292-1823

**Protocol Version (Date):** Amendment 1 (01 June 2016)

**Analysis Type:** Final

**Analysis Plan Version:** Version 1.0

**Analysis Plan Date:** 26 February 2018

Analysis Plan Author(s): PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

# **TABLE OF CONTENTS**

| TA | BLE O | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF I | N-TEXT TABLES | 4 |
| LIS | T OF A | ABBREVIATIONS | 5 |
| | | ODUCTION | |
| LIST C LIST C 1. IN 1. 1. 2. T 2. 3. G 3. 3. 3. 3. 3. 4. S 4. 5. B 5. 5. | | | |
| | 1.1.<br>1.2. | Study Objectives | |
| | 1.2. | Sample Size and Power | |
| 2 | | E OF PLANNED ANALYSIS | |
| 2. | | | |
| LIST 1. 2. 3. | 2.1. | Interim Analysis | |
| | 2.2. | 2.1.1. Week 24 AnalysisFinal Analysis | |
| | | • | |
| 3. | GEN. | ERAL CONSIDERATIONS FOR DATA ANALYSES | 10 |
| | 3.1. | Analysis Sets | |
| | | 3.1.1. All Randomized Analysis Set | |
| | | 3.1.2. Full Analysis Set | |
| | | 3.1.3. Safety Analysis Set | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates | |
| | 3.4. | Examination of Subject Subgroups | |
| | | 3.4.1. Subject Subgroups for Efficacy | |
| | 3.5. | 3.4.2. Subject Subgroups for Safety | |
| | 3.6. | Missing Data and Outliers | |
| | 3.0. | 3.6.1. Missing Data | |
| 1. In the state of | | 3.6.2. Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | |
| | 3.8. | Analysis Visit Windows | |
| | | 3.8.1. Definition of Study Day | |
| | | 3.8.2. Analysis Visit Windows | |
| LIST 1. I 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit | |
| | | Window | 16 |
| 4. | SUB | TECT DISPOSITION | 18 |
| | 4.1. | Subject Enrollment and Disposition. | 18 |
| | | 4.1.1. Subject Enrollment | |
| | | 4.1.2. Disposition of Subjects | |
| | 4.2. | Extent of Study Drug Exposure and Adherence | 19 |
| | | 4.2.1. Duration of Exposure to Study Drug | 19 |
| | | 4.2.2. Adherence to Study Drug | |
| | 4.3. | Protocol Deviations | 20 |
| 5. | BASI | ELINE CHARACTERISTICS | 21 |
| | 5.1. | Demographics | 21 |
| | 5.2. | Baseline Disease Characteristics | |
| | 5.3. | Medical History | |
| 6 | PPPI | CACY ANALYSES | |
| υ. | | | |

| | 6.1. | Primary | Efficacy Endpoint | 23 |
|---|---|---|---|---|
| | | 6.1.1. | Definition of Primary Efficacy Endpoint | 23 |
| | | 6.1.2. | US FDA-Defined Snapshot Algorithm | |
| | | 6.1.3. | Statistical Hypothesis for the Primary Efficacy Endpoint | |
| | | 6.1.4. | Primary Analysis of the Primary Efficacy Endpoint | |
| | 6.2. | | ary Efficacy Endpoints | |
| | | 6.2.1. | Definition of Secondary Efficacy Endpoints | |
| | | 6.2.2. | Analysis Methods for Secondary Efficacy Endpoints | |
| | 6.3. | | / Efficacy Endpoints | |
| | 0.5. | 6.3.1. | Definition of Tertiary Efficacy Endpoints | |
| | | 6.3.2. | Analysis of Tertiary Efficacy Endpoints | |
| | 6.4. | | s From Protocol-Specified Efficacy Analyses. | |
| _ | | Č | | |
| 7. | SAFE | TY ANA | LYSES | 29 |
| | 7.1. | Adverse | e Events and Deaths | |
| | | 7.1.1. | Adverse Event Dictionary | |
| | | 7.1.2. | Adverse Event Severity | 29 |
| | | 7.1.3. | Relationship of Adverse Events to Study Drug | 30 |
| | | 7.1.4. | Relationship of AEs to Study Procedure | 30 |
| | | 7.1.5. | Serious Adverse Events | |
| | | 7.1.6. | Treatment-Emergent Adverse Events | |
| | | 7.1.7. | Summaries of Adverse Events and Deaths | |
| | | 7.1.8. | Stage 3 Opportunistic Illnesses in HIV | |
| | | 7.1.9. | Potential Cardiovascular or Cerebrovascular Events | |
| | 7.2. | | ory Evaluations | |
| | 7.2. | 7.2.1. | Summaries of Numeric Laboratory Results | |
| | | 7.2.1. | Graded Laboratory Values | |
| | | 7.2.2. | Liver-Related Laboratory Evaluations | |
| | 7.3. | | afety Evaluations | |
| | 7.3. | 7.3.1. | • | |
| | | 7.3.1.<br>7.3.2. | Bone Biomarkers | |
| | 7.4 | , | Fracture Events | |
| | 7.4. | | afety Analyses | |
| | | 7.4.1. | Serum Creatinine | |
| | | 7.4.2. | Estimated Glomerular Filtration Rate | |
| | | 7.4.3. | Proteinuria by Urinalysis (Dipstick) | |
| | | 7.4.4. | Proteinuria by Quantitative Assessment | 38 |
| | | 7.4.5. | Urine Retinol Binding Protein to Creatinine Ratio and Beta-2- | |
| | | | Microglobulin to Creatinine Ratio | |
| | 7.5. | Vital Si | gns | 39 |
| | 7.6. | Prior an | nd Concomitant Medications | |
| | | 7.6.1. | Nonstudy-Drug Antiretroviral Medications | 39 |
| | | 7.6.2. | Concomitant Non-Antiretroviral Medications | 39 |
| | 7.7. | Electro | cardiogram Results | 40 |
| | 7.8. | Other S | afety Measures | 40 |
| | 7.9. | Change | s From Protocol-Specified Safety Analyses | 40 |
| 8. | PATI | ENT REP | ORTED OUTCOMES | 4 |
| | 8.1. | | nce – Visual Analogue Scale (VAS) Adherence Questionnaire | |
| | 0.1. | 8.1.1. | VAS Statistical Method | |
| | 8.2. | | VAS Statistical Method | |
| | 0.2. | ` | · | |
| | | 8.2.1. | Scoring the SF-36 | |
| | 0.2 | 8.2.2. | SF-36 Statistical Analysis Method | |
| | 8.3. | | eatment Satisfaction Questionnaire | |
| | | 8 3 1 | Scoring the HIV Treatment Satisfaction Questionnaire | 43 |

| | | 8.3.2. | HIV Treatment Satisfaction Questionnaire Statistical Analysis Method | 44 |
|---|---|---|---|---|
| | 8.4. | Function | al Assessment of Chronic Illness Therapy – Fatigue | |
| | | 8.4.1. | Scoring the Functional Assessment of Chronic Illness Therapy – Fatigue | 44 |
| | | 8.4.2. | Functional Assessment of Chronic Illness Therapy – Fatigue Analysis | |
| | | | Method | |
| | 8.5. | | 3L | |
| | | 8.5.1. | Scoring the EQ-5D-3L Descriptive System | |
| | | 8.5.2. | EQ-5D Single Summary Index | |
| | | 8.5.3. | Scoring the EQ VAS | |
| | | 8.5.4. | EQ-5D Statistical Analysis Method | 47 |
| 9. | REFE | RENCES . | | 48 |
| 10. | SOFT | WARE | | 49 |
| 11. | SAP F | REVISION | | 50 |
| 12. | A DDE | NDICEC | | 5. |
| 12. | APPE | NDICES | | 3 |
| | Apper | div 1 | Study Procedures Table | 51 |
| | Apper | | Flowchart of US FDA-Defined Snapshot Algorithm (for Switch Study Trial) | |
| | Apper | | Fracture Events | |
| | Apper | | Potential Cardiovascular or Cerebrovascular Events. | |
| | Apper | | UK TTO Value Set for EQ-5D-3L Questionnaire | |
| | Apper | | Medical History | |
| | Apper | | Programming Specification | |
| | пррег | idiri / . | 110g.unming openiculion | |
| | | | LIST OF IN-TEXT TABLES | |
| | Table | 3-1. | Analysis Visit Windows for HIV-1 RNA, CD4+ Cell Count, CD4%, Hematology, | |
| | | | Chemistry, Urinalysis and Urine Chemistry Laboratory Tests, eGFR <sub>CG</sub> , VAS, Vital | 1.4 |
| | Table | 2 2 | Signs and Weight Analysis Visit Windows for Evaluations of Bone and Renal Safety, HIVTSQs (at | 13 |
| | 1 abie | 3-2. | Day 1 Only) and HIVTSQc | 1.4 |
| | Table | 2 2 | Analysis Visit Windows for Fasting Glucose and Lipid Panels | |
| | Table | | Analysis Visit Windows for SF-36, FACIT-F, and EQ-5D-3L | |
| | Table | | Analysis Visit Windows for ECGs | |
| | Table | | List of Items on the HIVTSQ | |
| | Table | | Items by Subscale and Scoring Algorithm for FACIT-F | |
| | Table | | Computation of Aggregate Scores | |
| | Table | | Scores of EQ-5D-3L Descriptive System | |
| | Table | | Response Category for Responder Analysis | |
| | 1 4010 | 0 5. | response category for responder rularysis | |

#### LIST OF ABBREVIATIONS

3TC lamivudine
ABC abacavir
AE adverse event

ALP alkaline phosphatase
ALT alanine aminotransferase
ANOVA analysis of variance

ARV antiretroviral

AST aspartate aminotransferase

BMI body mass index
CI confidence interval

CMH Cochran-Mantel-Haenszel

COBI, /co cobicistat

CRF case report form
CSR clinical study report

DTG dolutegravir

E/C/F/TAF elvitegravir (EVG) 150 mg / cobicistat (COBI) 150 mg / emtricitabine (FTC) 200 mg /

tenofovir alafenamide (TAF) 10 mg single tablet regimen

ECG electrocardiogram

eGFR<sub>CG</sub> estimated glomerular filtration rate using Cockcroft-Gault formula

eGFR<sub>CKD-EPI, cvsC</sub> estimated glomerular filtration rate using CKD-EPI method based on serum cystatin C

ESDD early study drug discontinuation

ET early termination

FACIT-F Functional Assessment of Chronic Illness Therapy – Fatigue

FAS Full Analysis Set

FDA (United States) Food and Drug Administration

FDC fixed dose combination
GFR glomerular filtration rate

Gilead Gilead Sciences

HBcAb hepatitis B core antibody

HBsAg hepatitis B virus surface Antigen

HCVAb hepatitis C virus antibody

HCV hepatitis C virus

HIV human immunodeficiency virus

HIVTSQ HIV treatment satisfaction questionnaire

HLT high-level term

IWRS interactive web response system

LLT lower-level term
LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

PT preferred term

PTH parathyroid hormone

PVE pharmacovigilance and epidemiology

Q1, Q3 first quartile, third quartile RBP retinol binding protein

RPV rilpivirine RTV, /r ritonavir

SAP statistical analysis plan
SD standard deviation
SF-36 short form-36
SOC system organ class

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings

TTO time trade-off

ULN upper limit of normal

UACR urine albumin to creatinine ratio
UPCR urine protein to creatinine ratio

VAS visual analogue scale

WHO World Health Organization

## 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the clinical study report (CSR) for the final analysis for Study GS-US-292-1823. This SAP is based on the study protocol (Amendment 1) dated 01 June 2016 and the electronic case report form (eCRF). The SAP will be finalized prior to the data finalization date. Any changes made after the finalization of the SAP will be documented in the CSR.

#### 1.1. Study Objectives

The primary objective of this study is as follows:

To evaluate the efficacy of switching to E/C/F/TAF FDC relative to continuing on a baseline regimen consisting of ABC/3TC plus a third antiretroviral agent in maintaining HIV-1 RNA < 50 copies/mL at Week 24 (using FDA snapshot algorithm) in virologically suppressed, HIV-1 infected adult subjects</li>

The secondary objectives of this study are as follows:

- To evaluate the proportion of subjects maintaining virological response (defined as HIV-1 RNA < 50 copies/mL, FDA snapshot analysis) at Weeks 12 and 48
- To evaluate changes from baseline in CD4+ cell counts at Weeks 24 and 48
- To evaluate the safety and tolerability of the two treatment groups over 24 and 48 weeks

#### 1.2. Study Design

This is a randomized, open-label, multicenter study to evaluate the safety and efficacy of switching from ABC/3TC plus a third antiretroviral agent (as prescribed by the Investigator) to E/C/F/TAF FDC compared to staying on their current regimen in HIV-1 infected adult subjects who are virologically suppressed (HIV-1 RNA < 50 copies/mL) on a stable regimen containing ABC/3TC for  $\geq$  6 consecutive months prior to screening. Eligible subjects are randomly assigned to 1 of the following treatment groups in a 2:1 ratio:

- Treatment Group 1 (Immediate switch): Switch to E/C/F/TAF FDC (n = 200) at Day 1;
- Treatment Group 2 (Delayed switch): Continue on the current regimen of ABC/3TC plus a third antiretroviral agent for 24 weeks followed by a delayed switch to E/C/F/TAF FDC (n = 100).

Allowed third antiretroviral agents include:

| <b>Antiretroviral Class</b> | Agents |
|---|---|
| Boosted PI | ATV+COBI (or ATV/COBI FDC), DRV+COBI (or DRV/COBI FDC), DRV+RTV, LPV/r, ATV+RTV, FPV + RTV, SQV + RTV, ATV (no booster) |
| NNRTI | EFV, ETR, NVP, RPV |
| INSTI | DTG, RAL |

Central randomization is used. The randomization schedule is stratified by age group (< 60 years or  $\ge 60$  years).

The treatment duration is 48 weeks. After screening, eligible subjects will be randomized to immediate or delayed switch groups and treated for 48 weeks. Following the Screening and Day 1 visits, subjects will return for study visits at Weeks 4, 8, 12, 24, 36 and 48. Subjects randomized to the delayed switch group will also return for visits at Weeks 28 and 32.

Plasma HIV-1 RNA, laboratory analyses (CD4+ cell count, CD4%, serum chemistry, hematology, urinalysis and urine chemistry, estimated glomerular filtration rate (eGFR<sub>CG</sub>), pregnancy testing [for females of childbearing potential]), vital signs, weight, assessment of adverse events (AEs) and concomitant medications are performed at screening, baseline, Week 4, Week 8, Week 12, Week 24, Week 28 (delayed switch group only), Week 32 (delayed switch group only), Week 36, and Week 48/Early Study Drug Discontinuation (ESDD) visit.

Blood and urine for evaluation of bone and renal safety, inflammation and platelet and coagulation function are performed at baseline, Week 4, Week 12, Week 24, Week 28 (delayed switch group 2 only), Week 36 (delayed switch group only), and Week 48 visit.

Metabolic assessments are performed at baseline, Week 12, Week 24, Week 36 (delayed switch group 2 only), and Week 48.

12-Lead ECG (Performed Supine) is collected at screening and Week 48/ESDD only.

HBV and HCV serologies (ie, Hepatitis B virus surface Antigen [HBsAg], Hepatitis B core antibody [HBcAb], and Hepatitis C virus [HCVAb] serologies [reflex HCV RNA is performed in subjects with positive HCVAb serology]) are performed at screening only. Cystatin C and height are collected at screening only.

For further details of assessments taken at each visit, see Schedule of Assessments, Appendix 1.

#### 1.3. Sample Size and Power

With 200 subjects randomized to switch to the E/C/F/TAF FDC group at Day 1 and 100 subjects randomized to the delayed switch group at Week 24, the lower limit of the observed one sided 97.5% confidence interval will be expected to be greater than -0.120 (ie, non-inferiority margin of 12%) with > 90% power when the percentage of responders in both treatment groups for the primary endpoint is at least 90% at Week 24.

# 2. TYPE OF PLANNED ANALYSIS

# 2.1. Interim Analysis

# 2.1.1. Week 24 Analysis

Week 24 analysis was performed to assess the primary endpoint and the overall safety of the study cohort. The Week 24 analysis was performed after all subjects completed their Week 24 visit or prematurely discontinued from the study drug.

## 2.2. Final Analysis

The final analysis will be conducted after all subjects have completed the study or prematurely discontinued from the study.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (SD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

All statistical tests will be 2-sided and performed at the 5% significance level unless otherwise specified.

By-subject listings will be presented for all subjects in the All Randomized Analysis Set unless otherwise specified, and sorted by subject ID number, visit date, and time (if applicable). Data collected on log forms, such as AEs, will be presented in chronological order within subject. The treatment group to which subjects were randomized will be used in the listings.

In general, age (in years) on the date of the first dose of study drug will be used for analyses and presentation in listings. If a subject was not dosed with study drug, the date of randomization will be used instead of the first dose date of study drug. For screen failures, age on the date that informed consent was signed will be used.

Permanent discontinuation of study drug refers to premature discontinuation of study drug or completeness of study drug.

#### 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each table, figure, and listing. A summary of the number and percentage of subjects in each analysis set will be provided by the specified treatment group.

For analysis by treatment group, subjects will be grouped using the following terminology:

- Treatment Group 1: E/C/F/TAF;
- Treatment Group 2:
  - Up to Week 24: ABC/3TC+3rd Agent;
  - Post-Week 24: delayed switch to E/C/F/TAF.
- All E/C/F/TAF: all subjects who received at least one dose of study assigned E/C/F/TAF (both immediate and delayed switch to E/C/F/TAF).

Furthermore, for comparative summaries of safety data, only data through the Week 24 visit will be summarized and presented by treatment group (E/C/F/TAF and ABC/3TC + 3rd Agent).

# 3.1.1. All Randomized Analysis Set

The All Randomized Analysis set includes all subjects who are randomized into the study. This is the primary analysis set for by-subject listings.

## 3.1.2. Full Analysis Set

The Full Analysis Set (FAS) will include all the subjects who were randomized and received at least one dose of study drug (either E/C/F/TAF or ABC/3TC+3rd agent on or after Day 1). For the FAS, all efficacy data, including data collected after the last dose of study drug, will be included, unless specified otherwise. The FAS analysis set is the primary analysis set for the efficacy analyses.

#### 3.1.3. Safety Analysis Set

The Safety Analysis Set includes all randomized subjects who took at least 1 dose of E/C/F/TAF or ABC/3TC+3rd Agent (on or after Day 1). For subjects in Treament Group 1 and in Treatment Group 2 while on E/C/F/TAF, all data collected up to 30 days after subjects permanently discontinue study drug will be included in safety summaries, unless specified otherwise. For subjects in Treatment Group 2 while on ABC/3TC + 3rd Agent, all data collected up to the minimum of 30 days after subjects permanently discontinue study drug and 1 day prior to the start of E/C/F/TAF will be included in safety summaries, unless specified otherwise. This is the primary analysis set for safety analyses.

#### 3.2. Subject Grouping

For analyses based on the All Randomized Analysis Set or FAS, subjects will be grouped according to the treatment to which they were randomized. For analyses based on the safety analysis set, subjects will be grouped according to actual treatment received. The actual treatment received will be considered to be different from the randomized treatment only when the actual treatment differs from randomized treatment for the entire treatment duration.

#### 3.3. Strata and Covariates

Subjects will be randomly assigned to treatment groups via the the interactive web response system (IWRS) in a 2:1 allocation ratio using a stratified randomization schedule. Stratification will be based on the following variable:

• Age group (< 60 years or  $\ge 60$  years)

If there are discrepancies in stratification factor values between the IWRS and the clinical database, the values recorded in the clinical database will be used to stratify subjects for analyses.

## 3.4. Examination of Subject Subgroups

The stratification factor of age was used only to maintain balance between the treatment groups and is not considered a predictor or a prognostic factor for efficacy or safety.

## 3.4.1. Subject Subgroups for Efficacy

There are no prespecified subject subgroupings for efficacy analyses.

# 3.4.2. Subject Subgroups for Safety

There are no prespecified subject subgroupings for safety analyses.

#### 3.5. Multiple Comparisons

No prespecifed multiplicity adjustments are planned for confidence intervals and/or statistical tests.

## 3.6. Missing Data and Outliers

## 3.6.1. Missing Data

A missing datum for a given study visit window may be due to any of the following reasons:

- A visit occurred in the window but data were not collected or were unusable
- A visit did not occur in the window
- A subject permanently discontinued from the study before reaching the window.

In general, values for missing data will not be imputed, unless otherwise specified.

For missing last dosing date of study drug, imputation rules are described in Section 3.8.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.6.2, and for concomitant non-ARV medications in Section 7.6.2.

#### **3.6.2. Outliers**

Outliers will be identified during the data management and data analysis processes. All data will be included in the analyses. Unless specified otherwise, no sensitivity analyses to evaluate the impact of outliers on efficacy or safety outcomes are planned.

# 3.7. Data Handling Conventions and Transformations

Laboratory Data that are continuous in nature but are less than the lower limit of quantitation or above the upper limit of quantitation will be imputed as follows except for urine creatinine:

- A value that is 1 unit less than the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (x is considered as the limit of quantitation). For example, if the values are reported as < 20 and < 5.0, values of 19 and 4.9 will be used for calculation of summary statistics, respectively. An exception to this rule is: for values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used for calculation of summary statistics.
- A value that is 1 unit above the limit of quantitation will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (x is considered as the limit of quantitation). Values with decimal points will follow the same logic as above.
- The limit of quantitation will be used for calculation of descriptive statistics if the data is reported in the form of " $\leq$  x" or " $\geq$  x" (x is considered as the limit of quantitation).

For urine creatinine, value of "< 1" is handled as a missing value in its summary and the calculation of related ratios. HIV-1 RNA results of 'No HIV-1 RNA detected' and "<20 cp/mL HIV-1 RNA Detected" will be imputed as 19 copies/mL for analysis purposes. HCV RNA results of "<15 IU/mL HCV RNA detected" or "No HCV RNA detected" will be imputed as 14 IU/mL for analysis purposes.

#### 3.8. Analysis Visit Windows

## 3.8.1. Definition of Study Day

#### **Study Day 1:**

For subjects taking E/C/F/TAF, the date when the first dose of study drug was taken, as recorded on the Study Drug Administration eCRF form, will be used.

For subjects taking ABC/3TC+3rd Agent, the Day 1 visit date on the Visit Date eCRF will be used.

**Study Days** are calculated relative to Study Day 1. For events that occurred on or after Study Day 1 date, study days are calculated as (visit date minus Study Day 1 plus 1). For events that occurred prior to Study Day 1, study days are calculated as (visit date minus Study Day 1).

For subjects with delayed switch to E/C/F/TAF, the date when the first dose of E/C/F/TAF was taken, as recorded on the Study Drug Administration eCRF form, will be used as the first dose date for E/C/F/TAF.

#### Last Dose Date is defined as follows:

- For subjects taking E/C/F/TAF or delayed switch to E/C/F/TAF, the last dose date is defined as the latest of the study drug end dates recorded on the Study Drug Administration eCRF with "Permanently Withdrawn" box checked for subjects who prematurely discontinued or completed study drug according to the Study Drug Completion eCRF.
- For subjects taking ABC/3TC+3rd Agent who do not switch to E/C/F/TAF, the earliest stop date of any component (ie, ABC/3TC, or 3rd Agent, etc.) according to the Non-Study ARV Medication eCRF before switching to E/C/F/TAF or premature discontinuation will be used as the last dose date.
- For subjects taking ABC/3TC+3rd Agent who do switch to E/C/F/TAF, the last dose date of ABC/3TC+3rd Agent will be set as the day prior to the first dose date of E/C/F/TAF.

If the last dose date is missing or incomplete (eg, only year of last dose date is known or completely missing due to lost to follow-up) for subjects who prematurely discontinued study drug or completed the study drug, the latest of nonmissing study drug start dates and end dates, the clinical visit dates, and the laboratory visit dates, excluding the date of 30-day follow-up visit, will be used to impute the last dose date.

**Last Study Date** is the latest of nonmissing study drug start dates and end dates, the clinic visit dates, and the laboratory visit dates including the 30-day follow-up visit date for subjects who prematurely discontinued study or who completed study according to Study Completion eCRF.

**Baseline Value** is defined as the last nonmissing value obtained on or prior to Study Day 1 for HIV-1 RNA, CD4+ cell count, CD4%, hematology, chemistry, urinalysis and urine chemistry laboratory tests, fasting glucose and lipid panels, eGFR<sub>CG</sub>, cystatin C testing, vital signs and weight, safety electrocardiogram (ECG), Visual Analogue Scale (VAS) Adherence Questionnaire, SF-36 Questionnaire (SF-36), the HIV Treatment Satisfaction Questionnaire (HIVTSQ) – Status version (at Day 1 only), Functional Assessment of Chronic Illness Therapy – Fatigue (FACIT-F), and EQ-5D-3L.

#### 3.8.2. Analysis Visit Windows

Subject visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

In the description that follows, the column labelled "E/C/F/TAF" refers to subjects in the immediate and delayed switch group who have switched to E/C/F/TAF. The baseline for delayed switch subjects will be reset based on the date of first dose of E/C/F/TAF and the study day will be calculated relative to that date. Data collected after the date of switch to E/C/F/TAF will be excluded from the analysis of the ABC/3TC + 3rd Agent group.

The analysis windows for HIV-1 RNA, CD4+ cell count, CD4%, hematology, chemistry, urinalysis and urine chemistry laboratory tests, eGFR<sub>CG</sub>, VAS, vital signs and weight are provided in Table 3-1.

Table 3-1. Analysis Visit Windows for HIV-1 RNA, CD4+ Cell Count, CD4%, Hematology, Chemistry, Urinalysis and Urine Chemistry Laboratory Tests, eGFR<sub>CG</sub>, VAS, Vital Signs and Weight

| | | E/C/F/TAF | | ABC/3TC- | +3rd Agent |
|---|---|---|---|---|---|
| Nominal Visit | Nominal Day | Lower Limit | Upper Limit | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 | (none) | 1 |
| Week 4 | 28 | 2 | 42 | 2 | 42 |
| Week 8 | 56 | 43 | 70 | 43 | 70 |
| Week 12 | 84 | 71 | 126 | 71 | 126 |
| Week 24 | 168 | 127 | 210 | 127 | 210* |
| Week 36 | 252 | 211 | 294 | | |
| Week 48 | 336 | 295 | 420 | | |

<sup>\*</sup> For subjects who remained on study drug after Week 24, do not include data after the first dose date of E/C/F/TAF.

The analysis windows for evaluations of bone and renal safety (bone safety: parathyroid hormone [PTH] and serum OH-25 vitamin D; renal safety: retinol binding protein, and beta-2-microglobulin), HIVTSQs (at Day 1 only) and HIVTSQc are provided in Table 3-2.

Table 3-2. Analysis Visit Windows for Evaluations of Bone and Renal Safety, HIVTSQs (at Day 1 Only) and HIVTSQc

| | | E/C/F/TAF | | ABC/3TC- | +3rd Agent |
|---|---|---|---|---|---|
| Nominal Visit | Nominal Day | Lower Limit | Upper Limit | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 | (none) | 1 |
| Week 4 | 28 | 2 | 56 | 2 | 56 |
| Week 12 | 84 | 57 | 126 | 57 | 126 |
| Week 24 | 168 | 127 | 210 | 127 | 210* |
| Week 36 | 252 | 211 | 294 | | |
| Week 48 | 336 | 295 | 420 | | |

<sup>\*</sup> For subjects who remained on study drug after Week 24, do not include data after the first dose date of E/C/F/TAF.

The analysis windows for fasting glucose and lipid panels (including total cholesterol [TC], HDL, direct LDL, triglycerides, and TC to HDL ratio) are provided in the following table.

Table 3-3. Analysis Visit Windows for Fasting Glucose and Lipid Panels

| | | E/C/F/TAF | | ABC/3TC- | +3rd Agent |
|---|---|---|---|---|---|
| Nominal Visit | Nominal Day | Lower Limit | Upper Limit | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 | (none) | 1 |
| Week 12 | 84 | 2 | 126 | 2 | 126 |
| Week 24 | 168 | 127 | 252 | 127 | 252* |
| Week 48 | 336 | 253 | 420 | | |

<sup>\*</sup> For subjects who remained on study drug after Week 24, do not include data after the first dose date of E/C/F/TAF.

The analysis windows for SF-36, FACIT-F, and EQ-5D-3L are provided in the following table.

Table 3-4. Analysis Visit Windows for SF-36, FACIT-F, and EQ-5D-3L

| | | E/C/F/TAF | | ABC/3TC+3rd Agent | |
|---|---|---|---|---|---|
| Nominal Visit | Nominal Day | Lower Limit | Upper Limit | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 | (none) | 1 |
| Week 4 | 28 | 2 | 98 | 2 | 98 |
| Week 24 | 168 | 99 | 252 | 99 | 252* |
| Week 48 | 336 | 253 | 420 | | |

<sup>\*</sup> For subjects who remained on study drug after Week 24, do not include data after the first dose date of E/C/F/TAF.

The analysis windows for ECGs are provided in the following table.

Table 3-5. Analysis Visit Windows for ECGs

| | | E/C/F/TAF | | ABC/3TC- | +3rd Agent |
|---|---|---|---|---|---|
| Nominal Visit | Nominal Day | Lower Limit | Upper Limit | Lower Limit | Upper Limit |
| Baseline | 1 | (none) | 1 | (none) | 1 |
| Week 48 | 336 | 2 | (none) | 2 | (none)* |

<sup>\*</sup> For subjects who remained on study drug after Week 24, do not include data after the first dose date of E/C/F/TAF.

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require one value per analysis window. When a single value is needed, the following rule(s) will be used:

If multiple nonmissing numeric observations exist in a window, records will be chosen as follows:

- For baseline, the last available record on or prior to the date of the first dose of study drug will be selected. If there are multiple records with the same time or no time recorded on the same day, average will be used for the baseline value, except for HIV-1 RNA (see below).
- For postbaseline visits:
  - For CD4+ cell count, and CD4%, the record(s) collected on the latest day in the window will be selected for analysis.
  - For other numeric observations (ie, except HIV-1 RNA, CD4+ cell count, and CD4%), the record(s) collected on the day closest to the nominal day for that visit will be selected. If there are 2 days equidistant from the nominal day, the later day will be selected.
  - For any numeric observations except HIV-1 RNA, if there are multiple records on the selected day, the average will be taken.
- For baseline and postbaseline HIV-1 RNA, the latest (considering both date and time) record(s) in the window will be selected. If both "HIV RNA Taqman 2.0" and "HIV RNA Repeat" (ie, the HIV-1 RNA result obtained from an additional aliquot of the original sample) are available with the same collection time, the results from the "HIV RNA Repeat" will be selected for analysis purposes; otherwise, if there are multiple "HIV RNA Taqman 2.0" records with the same collection time, the geometric mean will be taken for analysis purposes.

If multiple valid nonmissing categorical observations (eg, safety ECG results) exist in a window, records will be chosen as follows:

- For baseline, the last available record on or prior to the date of the first dose of the study drug will be selected. If there are multiple records with the same time or no time recorded on the same day, the value with the lowest severity will be selected (eg, normal will be selected over abnormal for safety ECG findings).
- For postbaseline visits, the most conservative value within the window will be selected (eg, abnormal will be selected over normal for safety ECG)

#### 4. SUBJECT DISPOSITION

## 4.1. Subject Enrollment and Disposition

## 4.1.1. Subject Enrollment

The number and percentage of subjects randomized to each stratum (< 60 years or  $\ge$  60 years) will be summarized overall and by E/C/F/TAF and ABC/3TC+3rd Agent using the safety analysis set.

The number and percentage of subjects randomized in each country and by each investigator within a country will be summarized overall and by treatment group using the safety analysis set.

The enrollment related data will be listed. Subjects randomized to the incorrect stratum will be included in separate listing.

# 4.1.2. Disposition of Subjects

A summary of subject disposition will be provided overall and by E/C/F/TAF and ABC/3TC+3rd Agent. This summary will present the number and/or percentage of subjects screened, screen failure subjects who were not randomized, subjects who met all eligibility criteria and were not randomized, subjects randomized but not treated, subjects in the safety analysis set, subjects in the FAS set.

In addition, the number and percentage of subjects meeting the following criteria will be summarized by treatment group:

- Completed 24 weeks on randomized drug
- Switched to E/C/F/TAF (only for ABC/3TC + 3rd Agent subjects)
- Completed study drug
- Prematurely discontinued study drug (with summary of reasons for discontinuing study drug)
- Completed study
- Prematurely discontinued from the study (with summary of reasons for discontinuing the study).

The denominator for the percentage of subjects in each category will be the number of subjects in the safety analysis set.

No inferential statistics will be provided. A data listing of reasons for premature study drug discontinuation will be provided.

# 4.2. Extent of Study Drug Exposure and Adherence

Extent of exposure to study drug will be examined by assessing the total duration of exposure to study drug and the level of adherence to the study drug specified in the protocol. Adherence to study drug will be assessed only for subjects receiving E/C/F/TAF in the safety analysis set.

## 4.2.1. Duration of Exposure to Study Drug

Duration of exposure to study drug will be defined as (last dose date – first dose date + 1), regardless of temporary interruptions in study drug administration, and will be expressed in weeks (recorded to 1 decimal place, eg, 4.5 weeks). If the last dose date is not available, the latest of the study drug start dates and end dates, the clinical visit dates, and laboratory visit dates, excluding the 30-day follow-up visit date, will be used to impute the last dose date for the calculation of the duration of study drug exposure.

Duration of exposure to study drug will be summarized using descriptive statistics (n, mean, standard deviation [SD], median, Q1, Q3, minimum, and maximum). The number and percentage of subjects in the following categories will also be summarized:  $\geq 4$  weeks [28 days],  $\geq 8$  weeks [56 days],  $\geq 12$  weeks [84 days],  $\geq 24$  weeks [168 days],  $\geq 36$  weeks [252 days], and  $\geq 48$  weeks [336 days]. These categories start with a cumulative count thus subjects who complete the study will be counted from the first category up.

Summaries will be provided for subjects in the safety analysis set. No inferential statistics will be provided.

#### 4.2.2. Adherence to Study Drug

Study drug regimen adherence will be computed based on pill counts for exposure to E/C/F/TAF (both immediate and delayed switch groups). The numbers of pills of study drug (E/C/F/TAF) dispensed and returned are captured on Study Drug Accountability eCRF.

Adherence (%) of study drug regimen for E/C/F/TAF will be calculated as follows:

Adherence (%) = 100 
$$\times \frac{\text{Total Number of Pills Taken}}{\text{Total Number of Pills Prescribed}}$$

$$= 100 \times \frac{\sum \text{No. of pills taken at each dispensing period}^{[1]}}{\sum \text{No. of pills prescribed at each dispensing period}^{[2]}}$$

- [1] Number of pills taken at a distinct dispensing period for E/C/F/TAF is calculated as the minimum of (a) the daily number of pills prescribed for the study drug multiplied by **the duration of treatment** at the dispensing period of the same dispensing date, and (b) the number of pills taken for the study drug (number of pills dispensed minus the number of pills returned). Total number of pills taken is determined by summing the number of pills taken for the study drug from all evaluable dispensing periods.
- [2] Number of pills prescribed at a distinct dispensing period for a study drug is calculated as the daily number of pills prescribed for the study drug multiplied by the <u>duration of treatment</u> at the dispensing period of the same dispensing date. Total number of pills prescribed is determined by summing the number of pills prescribed for the study drug from all evaluable dispensing periods.

<u>The duration of treatment</u> at a dispensing period for a study drug is calculated as the minimum of (a) the last returned date of the same dispensing period for the study drug, (b) date of premature discontinuation of the study drug, and (c) <u>next pill dispensing date</u> of the study drug, minus dispensing date of the study drug.

<u>The next pill dispensing date</u> is the following dispensing date of the study drug regardless of the bottle return date.

For a record where the number of pills returned was missing (with "Yes" answered for "Was the Bottle returned?" question), it is assumed the number of pills returned was zero. If the number of pills dispensed was missing or any study drug bottle was not returned or the bottle return status was unknown, all records for the same dispensing date for that study drug will be excluded from both denominator and numerator calculation.

Overall adherence will be calculated for each subject for the entire dosing period up to the date of permanent discontinuation of the study drug for subjects who prematurely discontinued study drug.

Descriptive statistics for overall adherence and adherence up to Week 24 to study drug regimen (n, mean, SD, median, Q1, Q3, minimum and maximum) along with the number and percentage of subjects belonging to adherence categories (eg, < 80%,  $\ge 80\%$  to < 90%,  $\ge 90\%$  to < 95%,  $\ge 95\%$ ) will be provided for subjects receiving E/C/F/TAF in the safety analysis set for subjects who return at least 1 bottle and have calculable adherence during the study in the safety analysis set. No inferential statistics will be provided.

Adherence up to Week 24 visit will be calculated using all data from the entire dosing period up to the date of premature discontinuation of the study drug for subjects who prematurely discontinued study drug or completed study drug, or the Week 24 study drug dispensing date, whichever occurs earliest.

#### 4.3. Protocol Deviations

A listing will be provided for all randomized subjects who violated at least one inclusion or exclusion criterion. The listing will include the criteria not met. A listing of subjects who received the wrong study drug will also be provided.

## 5. BASELINE CHARACTERISTICS

## 5.1. Demographics

Subject demographic data (age, sex, race, and ethnicity) and baseline characteristics (body weight, height, body mass index [BMI]) will be summarized overall and by E/C/F/TAF and ABC/3TC+3rd Agent using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum and maximum) for continuous data and by the number and percent of subjects for categorical data. The summaries of demographic data and baseline characteristics will be provided using the safety analysis set. Age is calculated calculated as age in years at first dose of study drug.

For categorical data, the Cochran-Mantel-Haenszel (CMH) test (ie, general association statistic for nominal data) will be used to compare the 2 treatment groups. For continuous data, the 2-sided Wilcoxon rank sum test will be used to compare the 2 randomized treatment groups.

#### **5.2.** Baseline Disease Characteristics

The following baseline disease characteristics will be summarized overall and by E/C/F/TAF and ABC/3TC+3rd Agent:

- HIV-1 RNA categories (copies/mL): (a) < 50, (b)  $\ge 50$
- CD4+ cell count (/μL)
- CD4+ cell count categories (/ $\mu$ L): (a) < 50, (b)  $\geq$  50 to < 200, (c)  $\geq$  200 to < 350, (d)  $\geq$  350 to < 500, and (e)  $\geq$  500
- CD4 percentage (%)
- HIV risk factors (mode of infection): (a) Heterosexual Sex; (b) Homosexual Sex; (c) IV Drug Use; (d) Transfusion; (e) Vertical Transmission; (f) Other; (g) Unknown
- HIV disease status: (a) Asymptomatic; (b) Symptomatic HIV Infection; (c) AIDS
- HBV Surface Antigen Status (Negative/Positive)
- HCV Antibody Status (Negative/Positive/Indeterminate)
- Estimated GFR by CG (mL/min; see Section 7.4.2.1)
- Estimated GFR by CKD-EPI (mL/min; see Section 7.4.2.2)
- Proteinuria by urinalysis (dipstick; Negative/Trace/+1/+2/+3)

- Medical history: diabetes (Yes/No), hypertension (Yes/No), cardiovascular disease (Yes/No), and hyperlipidemia (Yes/No)
- Tobacco smoking history (Never Smoker/Former Smoker/Current Smoker)
- Genetic mother/father/ brother/sister with myocardial infarction/stroke before 50 years-old? (Yes/No/Unknown)
- Baseline ALT (U/L)
- Baseline AST (U/L)
- Baseline Platelet Count (10<sup>3</sup>/μL)
- ARV Regimen at Baseline

For categorical data (excluding HIV risk factors and ARV Regimen at Baseline), the Cochran-Mantel-Haenszel (CMH) test (general association statistic for nominal data and row means scores differ statistic for ordinal data) will be used to compare the 2 randomized treatment groups. For continuous data, a 2-sided Wilcoxon rank sum test will be used to compare the 2 randomized treatment groups.

A by-subject listing of baseline characteristics will be provided by subject ID number in ascending order.

# 5.3. Medical History

General medical history data will be collected at screening and listed only. General medical history data will not be coded.

# 6. EFFICACY ANALYSES

#### 6.1. Primary Efficacy Endpoint

## 6.1.1. Definition of Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 24 as defined by the FDA snapshot algorithm {U. S. Department of Health and Human Services 2015}. The proportions are expressed as percentages for presentation purpose.

## 6.1.2. US FDA-Defined Snapshot Algorithm

The analysis window at Week 24 is defined as from Study Day 127 to Study Day 210, inclusive. All HIV-1 RNA data collected on-treatment (ie, data collected up to 1 day after permanent discontinuation of study drug) will be used in the US FDA-defined snapshot algorithm. Virologic outcome will be defined as the following categories:

- **HIV-1 RNA < 50 copies/mL:** this includes subjects who have the last available on-treatment HIV-1 RNA < 50 copies/mL in the Week 24 analysis window
- HIV-1 RNA  $\geq$  50 copies/mL: this includes subjects:
  - 1) Who have the last available on-treatment HIV-1 RNA  $\geq$  50 copies/mL in the Week 24 analysis window while on randomized treatment, or
  - 2) Who do not have on-treatment HIV-1 RNA data in the Week 24 analysis window and
    - a) Who discontinue study drug prior to or in the Week 24 analysis window due to lack of efficacy (note: Lack of efficacy is defined as having the check-box for Lack of efficacy marked on the Study Drug Completion eCRF), or
    - b) Who discontinue study drug prior to or in the Week 24 analysis window due to AE or death and have the last available on-treatment HIV-1 RNA  $\geq$  50 copies/mL, or
    - c) Who discontinue study drug prior to or in the Week 24 analysis window due to reasons other than AE, death, or lack of efficacy and have the last available on-treatment HIV-1 RNA  $\geq$  50 copies/mL
- No Virologic Data (in the Week 24 Window): this includes subjects who do not have on-treatment HIV-1 RNA data in the Week 24 analysis window because of the following:
  - 1) Discontinuation of study drug prior to or in the Week 24 analysis window due to AE or death and the last available on-treatment HIV-1 RNA < 50 copies/mL, or
  - 2) Discontinuation of study drug prior to or in the Week 24 analysis window due to reasons other than AE, death, or lack of efficacy and the last available on-treatment HIV-1 RNA < 50 copies/mL, or
  - 3) Missing data during the window but on study drug.

The flowchart of snapshot algorithm is provided in Appendix 2.

Week 24 virologic outcomes for the US FDA-defined snapshot algorithm will also be listed.

*Note*: For switch study population, the US FDA-defined snapshot algorithm classifies subjects who discontinue study drug due to adverse event or death and have the last available on-treatment HIV-1 RNA value ≥ 50 copies/mL as HIV-1 RNA value ≥ 50 copies/mL. In the US FDA-defined snapshot algorithm for a treatment naïve study population, these subjects would be classified as having No Virologic Data in the Week 24 Analysis Window.

## 6.1.3. Statistical Hypothesis for the Primary Efficacy Endpoint

- **Null hypothesis:** E/C/F/TAF is at least 12% lower than the ABC/3TC+3rd Agent group with respect to the proportion of subjects with HIV-1 RNA < 50 copies/mL ("response rate") as determined by the FDA snapshot analysis at Week 24
- Alternative hypothesis: The E/C/F/TAF is less than 12% lower than the ABC/3TC+3rd Agent group with respect to the proportion of subjects with HIV-1 RNA < 50 copies/mL ("response rate") as determined by the FDA snapshot analysis at Week 24</li>

#### 6.1.4. Primary Analysis of the Primary Efficacy Endpoint

The analysis purpose of the primary efficacy endpoint is to assess the noninferiority of E/C/F/TAF relative to ABC/3TC+3rd Agent. Noninferiority will be assessed using an exact 2-sided 95% confidence interval (CI) based on an unconditional exact method using 2 inverted 1-sided tests with a noninferiority margin of 12% {Chan 1999}.

It will be concluded that E/C/F/TAF is non-inferior to ABC/3TC+3rd Agent if the lower bound of the 2-sided 95% CI of the difference in the response rate (E/C/F/TAF – ABC/3TC+3rd Agent) is greater than -12%. The primary analysis will use the FAS.

The number and percentage of subjects achieving HIV-1 RNA < 50 copies/mL, HIV-1 RNA ≥ 50 copies/mL, and reasons for no virologic data at Week 24 will be summarized.

If noninferiority of E/C/F/TAF versus ABC/3TC+3rd Agent is established, superiority of switching to E/C/F/TAF will be evaluated based on the same 95% CI used to evaluate noninferiority. If the lower bound of the 95% CI is greater than 0, then superiority of E/C/F/TAF over ABC/3TC+3rd Agent will be established. The 2-sided Fisher's exact test will also be used to assess superiority as a secondary assessment. The FAS set will be used for the superiority evaluation.

# 6.2. Secondary Efficacy Endpoints

## **6.2.1.** Definition of Secondary Efficacy Endpoints

Secondary efficacy endpoints are:

- Proportion of Subjects with HIV-1 RNA < 50 copies/mL at Weeks 12 and 48 as determined by US FDA-defined snapshot algorithm
- Proportion of subjects with HIV-1 RNA ≥ 50 copies/mL as defined by the US FDA-defined snapshot algorithm {U. S. Department of Health and Human Services 2015} at Weeks 12, 24, and 48.
- Change from baseline in CD4+ cell counts at Weeks 12, 24 and 48.

The analyses for the secondary efficacy endpoints will be conducted using the FAS analysis set.

## 6.2.2. Analysis Methods for Secondary Efficacy Endpoints

6.2.2.1. Analysis of Proportion of Subjects with HIV-1 RNA < 50 copies/mL as Defined by the US FDA-Defined Snapshot Algorithm at Week 12

The proportion of subjects with HIV-1 RNA < 50 copies/mL at Week 12 as determined by US FDA-defined snapshot algorithm will be analyzed similarly to the primary efficacy endpoint.

Similar to the primary efficacy endpoint, noninferiority will be assessed using the conventional CI approach. The point estimate of treatment difference (E/C/F/TAF – ABC/3TC+3rd Agent) in the percentage of subjects with HIV-1 RNA < 50 copies/mL and the associated 2-sided 95% CI will be constructed based on an unconditional exact method using 2 inverted 1-sided tests.

The above analysis will be performed using the full analysis set.

6.2.2.2. Analysis of Proportion of Subjects with HIV-1 RNA ≥ 50 copies/mL as Defined by the US FDA-Defined Snapshot Algorithm at Week 12 and 24

The proportion of subjects with HIV-1 RNA  $\geq$  50 copies/mL at Weeks 12 and 24 as determined by US FDA-defined snapshot algorithm will be analyzed similarly to the primary efficacy endpoint.

Similar to the primary efficacy endpoint, noninferiority will be assessed using the conventional CI approach. The point estimate of treatment difference (E/C/F/TAF – ABC/3TC+3rd Agent) in the percentage of subjects with HIV-1 RNA  $\geq$  50 copies/mL and the associated 2-sided 95% CI will be constructed based on an unconditional exact method using 2 inverted 1-sided tests.

The above analysis will be performed using the full analysis set.

6.2.2.3. Analysis of Proportion of Subjects with HIV-1 RNA < 50 copies/mL and ≥ 50 copies/mL as Defined by the US FDA-Defined Snapshot Algorithm at Week 48

The proportion of subjects with HIV-1 RNA < 50 copies/mL and  $\geq$  50 copies/mL at Week 48 as determined by US FDA-defined snapshot algorithm will be summarized descriptively for E/C/F/TAF subjects only using the full analysis set. No comparative statistics will be generated.

6.2.2.4. Analysis of CD4+ Cell Count at Weeks 12, 24, and 48

Analysis of CD4+ cell count will be based on on-treatment data using observed data (ie, missing will be excluded) for subjects in the FAS.

The change from baseline in CD4+ cell count at each scheduled visit will be summarized by E/C/F/TAF and ABC/3TC+3rd Agent using descriptive statistics.

The difference between treatment groups at baseline and change from baseline in CD4+ cell count between E/C/F/TAF and ABC/3TC+3rd Agent and the associated 95% CI will be constructed using analysis of variance (ANOVA) models including treatment as a fixed effect in the model through Week 24. P-values will be generated from the ANOVA model as well.

The mean and 95% CI of change from baseline in CD4+ cell count over time will be plotted for the FAS.

#### 6.3. Tertiary Efficacy Endpoints

#### 6.3.1. Definition of Tertiary Efficacy Endpoints

Tertiary efficacy endpoints are:

- The proportion of subjects with HIV-1 RNA < 20 copies/mL at Weeks 12, 24, and 48 as determined by the US FDA-defined snapshot algorithm. (See Section 6.1.2)
- The proportion of subjects with HIV-1 RNA < 50 copies/mL at Weeks 12, 24 and 48 as defined by 2 different missing data imputation methods.
- The change from baseline in CD4% at Weeks 12, 24 and 48.

The analyses for the tertiary efficacy endpoint will be conducted using the FAS.

# 6.3.2. Analysis of Tertiary Efficacy Endpoints

6.3.2.1. Analysis of Proportion of Subjects with HIV-1 RNA < 20 copies/mL at Weeks 12, 24, and 48 as Determined by the US FDA-Defined Snapshot Algorithm

The proportion of subjects with HIV-1 RNA < 20 copies/mL as determined by the US FDA-defined snapshot algorithm will be summarized at Weeks 12, 24, and 48 by E/C/F/TAF and ABC/3TC+3rd Agent using the same statistical methods specified in Sections 6.1.4, 6.2.2.1, and 6.2.2.3 above.

6.3.2.2. By Visit Summary of Proportion of Subjects with HIV-1 RNA < 50 copies/mL (Missing = Excluded and Missing = Failure Approaches)

The proportion of subjects with HIV-1 RNA < 50 copies/mL will also be analyzed by visit using the following 2 methods for imputing missing HIV-1 RNA values:

• Missing = Failure (M = F)

In this approach, all missing data will be treated as HIV-1 RNA  $\geq$  50 copies/mL. The denominator for percentages at a visit is based on the number of subjects in the FAS.

• Missing = Excluded (M = E)

In this approach, all missing data will be excluded in the computation of the proportions (ie, missing data points will be excluded from both the numerator and denominator). The denominator for percentages at a visit is based on the number of subjects in the FAS with non-missing HIV-1 RNA value at that visit.

For both M = F and M = E analyses, the number and percentage of subjects with HIV-1 RNA in the following categories will be summarized by visit:

- < 50 copies/mL
- < 20 copies/mL
  - < 20 copies/mL Not Detectable
  - < 20 copies/mL Detectable
- 20 to < 50 copies/mL
- 50 to < 200 copies/mL
- 200 to < 400 copies/mL
- 400 to < 1000 copies/mL

- $\geq 1000 \text{ copies/mL}$
- Missing (only applicable for M = F analysis)

For M = F analysis, results will be summarized and plotted by E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF for all visits. For M = E analysis, results will be summarized by E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF for all visits. The same statistical methods as applied to the analysis of the US FDA-defined snapshot algorithm will be used.

## 6.3.2.3. Analysis of CD4% at Weeks 12 and 24

Analysis of CD4% will be based on on-treatment data.

The difference between treatment groups at baseline and change from baseline in CD4% at each scheduled visit will be summarized by E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics.

The difference in change from baseline in CD4% between E/C/F/TAF and ABC/3TC+3rd Agent and the associated 95% CI will be constructed using ANOVA models including treatment as a fixed effect in the model through Week 24. P-values will be generated from the ANOVA model as well.

# 6.4. Changes From Protocol-Specified Efficacy Analyses

No change from the protocol-specified efficacy analysis is planned.

#### 7. SAFETY ANALYSES

Safety data will be summarized for the subjects in the safety analysis set. All safety data collected up to 30 days after permanent discontinuation of study drug will be summarized by treatment group, unless specified otherwise. All safety data will be included in data listings.

#### 7.1. Adverse Events and Deaths

Summaries of AEs will include data collected up to:

- for subjects randomized to or had switched to E/C/F/TAF and have permanently discontinued study drug, the last dose of study drug plus 30 days.
- for subjects randomized to ABC/3TC+3rd Agent and were receiving ABC/3TC+3rd Agent, the minimum of (1) 30 days after permanent discontinuation of ABC/3TC+3rd Agent or (2) the first dose date of E/C/F/TAF 1 (AEs and concomitant medications) will be summarized, unless specified otherwise.

Summaries of AEs up to Week 24 will include data collected up to:

- for subjects randomized to E/C/F/TAF, the minimum of (1) 30 days after permanent discontinuation of study drug or (2) the Week 24 visit.
- for subjects randomized to ABC/3TC+3rd Agent, the minimum of (1) 30 days after permanent discontinuation of ABC/3TC+3rd Agent or (2) the first dose date of E/C/F/TAF 1 (AEs and concomitant medications) will be summarized, unless specified otherwise.

All AEs analysis described below will be repeated using adverse events up to Week 24. Analyses up to Week 24 will be summarized by E/C/F/TAF and ABC/3TC+3rd Agent only.

#### 7.1.1. Adverse Event Dictionary

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, latest version). System organ class (SOC), high level group term (HLGT), high level term (HLT), preferred term (PT), and lowest-level term (LLT) will be attached to the clinical database.

## 7.1.2. Adverse Event Severity

AEs are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) or Grade 4 (life threatening) according to toxicity criteria specified in the study Protocol Appendix 4. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings, and will be considered the least severe for the purposes of sorting for data presentation.

# 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator answers "Related" to the question "Related to Study Treatment?" in the CRF. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show relationship as missing.

## 7.1.4. Relationship of AEs to Study Procedure

Adverse events for which "Yes" is marked for question "Related to Study Procedures?" in the eCRF will be identified and included in the AE listing.

#### 7.1.5. Serious Adverse Events

Serious adverse events (SAEs) are those identified as serious in the clinical database. The clinical database will be reconciled with the SAE database from the Pharmacovigilance and Epidemiology (PVE) Department before database finalization.

# 7.1.6. Treatment-Emergent Adverse Events

#### 7.1.6.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

For subjects randomized to or had switched to E/C/F/TAF:

- any AE with onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug, or
- any AE leading to premature discontinuation of study drug.

For subjects randomized to ABC/3TC+3rd Agent and were receiving ABC/3TC+3rd Agent:

- any AE with onset date on or after the ABC/3TC+3rd Agent first dose date and the minimum of (1) the last dose date of ABC/3TC+3rd Agent plus 30 days and (2) the first dose date of E/C/F/TAF 1 or
- any AE leading to premature discontinuation of ABC/3TC and/or 3rd Agent.

#### 7.1.6.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent if both of the following 2 criteria are met:

- The month and year of the AE onset date is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The month and year of the AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the date of the last dose of study drug

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date marked as ongoing or on or after the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

#### 7.1.7. Summaries of Adverse Events and Deaths

A brief summary of AEs will show, by treatment group, the number and percentage of subjects who (1) had any treatment-emergent AE, (2) had any Grade 3 or 4 treatment-emergent AE, (3) had any Grade 2, 3, or 4 treatment-emergent AE, (4) had any treatment-emergent study drug-related AE, (5) had any Grade 3 or 4 treatment-emergent study drug-related AE, (6) had any Grade 2, 3, or 4 treatment-emergent study drug-related AE, (7) had any treatment-emergent SAE, (8) had any treatment-emergent study drug-related SAE, (9) had any treatment-emergent AE leading to premature study drug discontinuation, and (10) had treatment-emergent death. Treatment-emergent death refers to death occurring between the first dose date and the last dose date plus 30 days (inclusive).

Summaries (number and percentage of subjects) of AEs (by SOC, HLT [if specified below], and PT) will be provided for E/C/F/TAF, ABC/3TC+3rd Agent, delayed switch to E/C/F/TAF, and All E/C/F/TAF using the safety analysis set as follows:

- All TEAEs summarized by SOC, HLT, and PT
- Any Grade 3 or 4 TEAEs
- Any Grade 2, 3, or 4 treatment-emergent AEs
- All treatment-emergent study drug-related AEs
- All Grade 3 or 4 treatment-emergent study drug-related AEs
- Any Grade 2, 3, or 4 treatment-emergent study drug-related AEs
- All treatment-emergent serious AEs
- All treatment-emergent study drug-related SAEs
- All treatment-emergent AEs leading to premature discontinuation of study drug

Multiple events will be counted only once per subject in each summary. For data presentation, SOC (and HLT) will be ordered alphabetically, with PT sorted by decreasing total frequency. For summaries by severity grade, the most severe event will be selected.

In addition to the above summary tables, all TEAEs and TE study drug-related AEs will be summarized by PT only, in descending order of total frequency.

A second set of summaries will be produced that only summarizes E/C/F/TAF and ABC/3TC + 3rd Agent through the Week 24 visit.

Data listings will be provided for the following:

- All AEs
- Grade 3 and 4 AEs
- SAEs
- Study Drug-Related SAEs
- Deaths
- Adverse events leading to premature discontinuation of study drug

## 7.1.8. Stage 3 Opportunistic Illnesses in HIV

On an ongoing basis, AEs will be reviewed for events that might meet the definition of stage 3 opportunistic illnesses in HIV that are indicative of an AIDS-Defining Diagnoses (see Protocol Appendix 6). The Gilead medical monitor will review the possible stage 3 opportunistic illnesses and approve the events that meet the definition. Events that meet the stage 3 opportunistic illness definition of an AIDS-Defining Diagnosis will be listed.

#### 7.1.9. Potential Cardiovascular or Cerebrovascular Events

Potential cardiovascular or cerebrovascular events are defined as events coded to the PT in the selected PT listing, which was provided by Gilead PVE and reviewed by Gilead medical monitors (see Appendix 4).

A summary (number and percentage of subjects) of potential treatment-emergent cardiovascular or cerebrovascular events by PT will be provided by treatment group (including the All E/C/F/TAF group) based on the safety analysis set. A second summary will be prepared that only includes E/C/F/TAF and ABC/3TC+3rd Agent (up to Week 24). The second summary will contain a statistical comparison of the subject incidence rates (up to Week 24) between E/C/F/TAF and ABC/3TC+3rd Agent using Fisher's exact test. A data listing of potential cardiovascular or cerebrovascular events will be provided.

#### 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the safety analysis set and will include data collected up to:

- for subjects randomized to or had switched to E/C/F/TAF, and have permanently discontinued study drug, the last dose of study drug plus 30 days.
- for subjects randomized to ABC/3TC+3rd Agent and were receiving ABC/3TC+3rd Agent, the minimum of (1) the last dose date of ABC/3TC+3rd Agent plus 30 days or (2) the first dose date of E/C/F/TAF.

The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7.

A by-subject listing for laboratory test results will be provided by subject ID number and visit in chronological order for hematology, serum chemistry, and urinalysis separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the Gilead Grading Scale for Severity of Adverse Events and Laboratory Abnormalities will be flagged in the data listings, as appropriate.

## 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics (n, mean, standard deviation, median, Q1, Q3, minimum and maximum) will be provided for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF for each laboratory test specified in the study protocol as follows:

- Baseline values
- Values at each postbaseline analysis window
- Change from baseline to each postbaseline analysis window
- Percentage change from baseline to each postbaseline analysis window (if specified)

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

#### 7.2.1.1. Metabolic Assessments

For the metabolic assessments (including total cholesterol, low density lipoprotein [LDL], high density lipoprotein [HDL], total cholesterol to HDL ratio, triglycerides, and glucose), only those measurements under fasting status will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF. P-values for the difference between E/C/F/TAF and ABC/3TC+3rd Agent in baseline and postbaseline values as well as the change from baseline (up to Week 24) in metabolic assessment will be estimated from the 2-sided Wilcoxon rank sum test to compare E/C/F/TAF and ABC/3TC+3rd Agent.

In addition, the number and percentage of subjects who took lipid modifying medications at the study entry and initiated the medications during the study (up to Week 24) will be provided, respectively. Statistical comparisons of the subject incidence rates between E/C/F/TAF and ABC/3TC+3rd Agent will be performed using Fisher's exact test.

A lipid modifying medication is defined as a medication with drug class = "LIPID MODIFYING AGENTS" and CMDECOD containing the wording of "STATIN".

A sensitivity analysis of fasting lipid tests (including total cholesterol, LDL, HDL, triglycerides, and total cholesterol to HDL ratio) will be performed by excluding subjects who took lipid modifying medications at study entry or initiated the medications during the study: baseline, and Week 24 and changes from baseline at Week 24 will be summarized by E/C/F/TAF and ABC/3TC+3rd Agent and p-values for the difference between E/C/F/TAF and ABC/3TC+3rd Agent will be estimated from a 2-sided Wilcoxon rank sum test. Only subjects with both baseline and Week 24 values will be included in the analysis.

Median (Q1, Q3) change from baseline in fasting metabolic assessments over time will be plotted for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF.

#### 7.2.1.2. Calcium Corrected for Albumin

Calcium corrected for albumin will be calculated and summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF. The following formula will be used when both serum calcium and albumin results for a given blood draw are available and serum albumin value is < 4.0 g/dL.

Calcium corrected for albumin (mg/dL) = serum calcium (mg/dL) +  $0.8 \times (4.0 - \text{albumin (g/dL)})$ . Toxicity grading for calcium will be applied based on the corrected values.

## 7.2.2. Graded Laboratory Values

The criteria specified in the study protocol will be used to grade laboratory results as Grade 0, mild (Grade 1), moderate (Grade 2), severe (Grade 3) or potentially life threatening (Grade 4). Grade 0 includes all values that do not meet criteria for an abnormality of at least Grade 1. Some laboratory tests have criteria for both increased and decreased levels; analyses for each direction (i.e., increased, decreased) will be presented separately.

For triglycerides, LDL, and cholesterol, the protocol specified toxicity grade scale is for fasting test values, so nonfasting lipid results (or lipid results without known fasting status) will not be graded or summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF by toxicity grades.

If there is any laboratory toxicity grading scale overlapping with normal reference ranges (eg, Grade 1 scale overlaps with normal reference ranges), laboratory values within normal range will be grade 0, except lipid tests.

## 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least one toxicity grade from baseline at any time post-baseline up to the cutoffs specified at the start of Section 7.2.

If the relevant baseline laboratory data are missing, then any abnormality of at least Grade 1 will be considered treatment emergent.

Serum glucose, fasting glucose and nonfasting glucose (including glucose results without a known fasting status) are graded based on different grading criteria as specified in the protocol. Treatment-emergent laboratory abnormalities will be summarized for fasting glucose. Since nonfasting glucose was not assessed at baseline, the maximum postbaseline grade instead of treatment-emergent laboratory abnormalities will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF.

#### 7.2.2.2. Summaries of Laboratory Abnormalities

The following summaries (number and percentage of subjects) of laboratory abnormalities will be provided for E/C/F/TAF, ABC/3TC+3rd Agent, delayed switch to E/C/F/TAF and All E/C/F/TAF (categorized according to most severe abnormality grade):

- Treatment-emergent laboratory abnormalities
- Treatment-emergent Grade 3 and 4 laboratory abnormalities

A second set of summaries will be produced that only summarizes E/C/F/TAF and ABC/3TC + 3rd Agent through the Week 24 visit.

For all summaries of laboratory abnormalities, the denominator is the number of subjects with non-missing post-baseline values for the lab test, obtained up to 30 days after permanent discontinuation of study drug. A listing of all graded laboratory abnormalities and all Grade 3 or Grade 4 laboratory abnormalities will be provided.

# 7.2.3. Liver-Related Laboratory Evaluations

The number and percentage of subjects will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, delayed switch to E/C/F/TAF, and All E/C/F/TAF for the following liver-related laboratory tests and categories:

- Aspartate aminotransferase (AST): (a) > 3 x Upper limit of normal (ULN), (b) > 5 x ULN,
   (c) > 10 x ULN, (d) > 20 x ULN
- Alanine aminotransferase (ALT): (a) > 3 x ULN, (b) > 5 x ULN, (c) > 10 x ULN,
   (d) > 20 x ULN
- AST or ALT: (a) > 3 x ULN, (b) > 5 x ULN, (c) > 10 x ULN, (d) > 20 x ULN
- Total bilirubin: (a)  $> 1 \times ULN$ , (b)  $> 2 \times ULN$
- Alkaline phosphatase (ALP) > 1.5 x ULN
- AST or ALT > 3 x ULN and total bilirubin: (a) > 1.5 x ULN, (b) > 2 x ULN
- AST or ALT > 3 x ULN and total bilirubin > 2 x ULN and ALP < 2 x ULN

For individual laboratory tests, subjects will be counted once based on the most severe postbaseline values. For both the composite endpoint of AST or ALT and total bilirubin, and the composite endpoint of AST or ALT, total bilirubin, and ALP, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the safety analysis set with nonmissing postbaseline value of the tests in evaluation at the same postbaseline visit date.

A second summary will be produced that only summarizes E/C/F/TAF and ABC/3TC + 3rd Agent through the Week 24 visit.

Subjects with AST or ALT > 3 x ULN will also be listed.

#### 7.3. Bone Safety Evaluations

#### 7.3.1. Bone Biomarkers

Bone safety evaluations include parathyroid (PTH) and serum OH-25 vitamin D.

Baseline, postbaseline, change from baseline, and percentage change from baseline in bone safety evaluations at each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics. The difference in percentage change from baseline (through Week 24) in these parameters between E/C/F/TAF and ABC/3TC+3rd Agent will be tested using a 2-sided Wilcoxon rank sum test.

Median (Q1, Q3) percentage change from baseline in bone safety evaluations over time will be plotted for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF. A listing of bone biomarker data will be provided.

#### 7.3.2. Fracture Events

The PTs for fracture events were defined based on Standardised MedDRA Query (SMQ) of Osteoporosis/Osteopenia. Fracture events will be summarized based on the identified PTs from SMQ. The number and percentage of subjects who experienced fracture events will be provided by treatment group (including the All E/C/F/TAF group) based on the safety analysis set. A second summary will be prepared that only includes E/C/F/TAF and ABC/3TC+3rd Agent (up to Week 24). The second summary will contain a statistical comparison of the subject incidence rates (up to Week 24) between E/C/F/TAF and ABC/3TC+3rd Agent using Fisher's exact test.

A data listing of fracture events will be provided.

#### 7.4. Renal Safety Analyses

#### 7.4.1. Serum Creatinine

The baseline, postbaseline and change from baseline in serum creatinine at each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics. Differences in baseline, postbaseline, and change from baseline between E/C/F/TAF and ABC/3TC+3rd Agent at each study visit (through Week 24) will be assessed
using a 2-sided Wilcoxon rank-sum test. A second set of summaries will be generated in subjects receiving (as well as not receiving) a creatinine secretion inhibitor at baseline (defined as having a baseline ARV regimen consisting of any of the following: cobicistat [appearing as "/co"], dolutegravir [appearing as "DTG"], rilpivirine [appearing as "RPV"], or ritonavir [appearing as either "RTV" or "/r"]).

Median (Q1, Q3) change from baseline in observed serum creatinine over time will be plotted for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF.

#### 7.4.2. Estimated Glomerular Filtration Rate

#### 7.4.2.1. Estimated Glomerular Filtration Rate: Cockcroft-Gault

The Cockcroft-Gault formula will be used to calculate eGFR<sub>CG</sub>:

$$eGFR_{CG}$$
 (mL/min) = [(140 – age (years)) × weight (kg) × (0.85 if female)] / (SCr (mg/dL) × 72),

where weight is total body mass in kilograms, and SCr is serum creatinine.

Summary of baseline, post-baseline, and change from baseline in eGFR<sub>CG</sub> at each visit will be provided for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF. Differences in baseline, postbaseline, and change from baseline between E/C/F/TAF and ABC/3TC+3rd Agent at each study visit (through Week 24) will be assessed using a 2-sided Wilcoxon rank-sum test. A second set of summaries will be generated in subjects receiving (as well as not receiving) a creatinine secretion inhibitor at baseline, defined above.

Median (Q1, Q3) change from baseline in eGFR<sub>CG</sub> over time will be plotted for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF.

#### 7.4.2.2. Estimated Glomerular Filtration Rate: CKD-EPI (cystatin C)

The CKD-EPI (cystatin C) formula will be used to calculate eGFR<sub>CKD-EPI, cysC</sub>:

eGFR<sub>CKD-EPI</sub> (mL/min/1.73 m<sup>2</sup>) =  $133 \times min(Scys/0.8, 1)^{-0.499} \times max(Scys/0.8, 1)^{-1.328} \times 0.996^{Age}$  [× 0.932 if female],

where Scys is serum cystatin C (mg/L), min (Scys/0.8,1) indicates the minimum of Scys/0.8 or 1, and max (Scys/0.8,1) indicates the maximum of Scys/0.8 or 1.

Only baseline values will be summarized. See Section 5.2 for details. Differences at baseline between E/C/F/TAF and ABC/3TC+3rd Agent will be assessed using a 2-sided Wilcoxon rank-sum test.

## 7.4.3. Proteinuria by Urinalysis (Dipstick)

The proteinuria by urinalysis (dipstick) toxicity grade (Grade 0 to Grade 3) at Weeks 12 and 24, will be summarized by baseline proteinuria toxicity grade for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF. In addition, the last on-treatment (ie, data collected up to 1 day after permanent discontinuation the last dose date of study drug) proteinuria toxicity grade will also be summarized by baseline proteinuria toxicity grade and treatment group.

The distribution of proteinuria toxicity grade at Weeks 12 and 24 and at the last on-treatment value, respectively, will be compared between E/C/F/TAF and ABC/3TC+3rd Agent adjusting for baseline proteinuria toxicity grade using rank analysis of covariance {LaVange 2008}.

## 7.4.4. Proteinuria by Quantitative Assessment

The baseline, postbaseline, changes from baseline, and percentage change from baseline in urine protein to creatinine ratio (UPCR) and urine albumin to creatinine ratio (UACR) at each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics. Differences in baseline and percent change from baseline between E/C/F/TAF and ABC/3TC+3rd Agent at each study visit (through Week 24) will be assessed using a 2-sided Wilcoxon rank-sum test.

The number and percentage of subjects with UPCR  $\leq$  200 mg/g versus > 200 mg/g will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF by baseline category at Week 24, and based on the last on-treatment value.

The number and percentage of subjects with UACR < 30 mg/g versus  $\ge 30$  mg/g will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF by baseline category at Week 24, and the last on-treatment value.

Median (Q1, Q3) percentage change from baseline in UPCR and UACR over time will be plotted for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF.

# 7.4.5. Urine Retinol Binding Protein to Creatinine Ratio and Beta-2-Microglobulin to Creatinine Ratio

Renal safety evaluations include urine retinol binding protein (RBP) to creatinine ratio and beta-2-microglobulin to creatinine ratio.

Baseline, postbaseline, change from baseline, and percentage change from baseline in urine RBP to creatinine ratio and beta-2-microglobulin to creatinine ratio at each visit will be summarized using descriptive statistics. Differences in baseline and percent change from baseline between E/C/F/TAF and ABC/3TC+3rd Agent at each study visit (through Week 24) will be assessed using a 2-sided Wilcoxon rank-sum test.

Median (Q1, Q3) percent change from baseline in urine RBP to creatinine ratio and beta-2-microglobulin to creatinine ratio over time will be plotted by treatment group.

## 7.5. Vital Signs

Descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) at each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF as follows:

- Baseline values
- Values at each postbaseline analysis window
- Change from baseline to each postbaseline analysis window

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

A listing of weight, BMI, height, and vital signs will be provided.

#### 7.6. Prior and Concomitant Medications

#### 7.6.1. Nonstudy-Drug Antiretroviral Medications

Nonstudy drug ARV medications used prior to, during, or after the study (if collected), will be coded using the GSI-modified WHO Drug Dictionary. The WHO preferred name and drug code will be attached to the clinical database. All nonstudy-drug ARV medications will be listed. No inferential statistics will be provided.

#### 7.6.2. Concomitant Non-Antiretroviral Medications

Concomitant non-ARV medications (ie, medications other than study drug that are taken while receiving study drug) will be coded using the WHO Drug Dictionary. The WHO preferred name and drug code will be attached to the clinical database. Use of concomitant medications will be summarized (number and percentage of subjects) by WHO drug class and preferred name for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF. Multiple drug use (by preferred name) will be counted once only per subject. The summary will be sorted alphabetically by drug class and then by decreasing total frequency within a class.

Non-ARV medications are defined as concomitant if:

- for subjects randomized to or had switched to E/C/F/TAF, they are taken from date of the first dose of study drug up to the date of the last dose of study drug;
- for subjects randomized to ABC/3TC+3rd Agent and were receiving ABC/3TC+3rd Agent, they are taken from the baseline visit date up to the last dose date as defined in Section 3.8.1.

If the start or stop date of non-ARV medications is incomplete, the month and year (or year alone if month is not recorded) of start or stop date will be used to determine whether the non-ARV medications are concomitant or not as follows. The medication is concomitant if the month and year of start or stop (or year of the start or stop) of the medication do not meet any of following criteria:

- The month and year of start of the medication is after the date of the last dose of study drug
- The month and year of stop of the medication is before the date of the first dose of study drug

If the start and stop date of non-ARV medications are not missing, the start date is not after last dose date and the stop date is not before first dose date, or the non-ARV medications are marked as ongoing and start date is on or before last dose date, the non-ARV medications are concomitant.

Summaries of concomitant non-ARV medications will be provided for the safety analysis set. Subjects with any concomitant non-ARV medications will be listed. No inferential statistics will be provided.

#### 7.7. Electrocardiogram Results

A listing of safety ECG results will be provided including treatment, assessment date and time, and ECG results.

#### 7.8. Other Safety Measures

A data listing will be provided for subjects experiencing pregnancy during the study.

### 7.9. Changes From Protocol-Specified Safety Analyses

The protocol specified that Safety ECGs will be listed and summarized for subjects in the Safety Analysis Set. However, subjects in Treatment Arm 2 do not have any postbaseline assessments while on ABC/3TC + 3rd agent. As such, safety ECG results will only be listed.

#### 8. PATIENT REPORTED OUTCOMES

The Patient reported outcomes (PROs) include: (1) Visual Analogue Scale (VAS) adherence questionnaires; (2) Short Form-36 Version 2 Health Survey (SF-36); (3) HIVTSQ (Status version at Day 1 only and Change version for other visits); (4) FACIT-F; (5) EQ-5D-3L.

PRO data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries will be provided for the safety analysis set and will include data:

- for subjects randomized to or had switched to E/C/F/TAF, and have permanently discontinued study drug, all data collected up to the last dose of study drug plus 30 days.
- for subjects randomized to ABC/3TC+3rd Agent and were receiving ABC/3TC+3rd Agent, all data collected up to the minimum of (1) the last dose date of ABC/3TC+3rd Agent plus 30 days or (2) the first dose date of E/C/F/TAF.

Unless otherwise stated, multiple responses and out of range responses will be set to missing and missing responses will not be imputed. The safety analysis set will be used in all analyses. All reported data will be listed.

### 8.1. Adherence – Visual Analogue Scale (VAS) Adherence Questionnaire

The visual analogue scale (VAS) adherence questionnaire is a 3-item, self-reported questionnaire that assesses the degree to which ARV medication was taken in the past 30 days.

For the VAS, the subject is asked to describe their adherence to their ARV regimen by using a linear scale (0% - 100%) to indicate what percent of medications was taken in the last 30 days (0% = taken none of prescribed anti-HIV medication), and 100% = taken all doses of prescribed anti-HIV medication). Two additional questions ask how many days the subject has missed medications in the last 30 days and how many days the subject has missed medications in the last 4 days.

#### 8.1.1. VAS Statistical Method

The VAS (%) absolute value and its change from baseline at each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics. The 2-sided Wilcoxon rank-sum test will be used to compare the difference between E/C/F/TAF and ABC/3TC+3rd Agent at baseline and in the change from baseline at each visit (through Week 24).

Number of days with missed doses in the past 30 days and past 4 days will be summarized categorically (eg, < 2, 2 to < 4, 4 to < 6,  $\ge 6$  for the past 30 days; 0 and > 0 for the past 4 days) at each visit

## 8.2. SF-36 (Version 2) Health Survey

The SF-36 Version 2 is a 36-item, self-reported, generic, comprehensive, and widely used questionnaire that is designed to measure health-related quality of life in the general population, as well as in subject groups with diverse chronic diseases including HIV/AIDS. Responses from the 36 items are used to construct 8 health domains including physical functioning, social functioning, general health, vitality, bodily pain, mental health, role capacity-physical, and role capacity-emotional. Furthermore, 2 summary scores, the Physical Component Summary (PCS) score and Mental Component Summary (MCS) score, aggregate information from the 8 SF-36 domains in a way that captures 80% to 85% of the variance in the 8 domains.

## 8.2.1. Scoring the SF-36

The 8 domains and 2 component summary scores of the SF-36 will be calculated according to "How to Score Version 2 of the SF-36 Health Survey (Chapters 6 and 7)" {Maruish 2011} published by QualityMetric Inc using 2009 population norms. Scores for each of the 8 domain including PCS and MCS range from 0 to 100 with higher score indicating better functioning.

## 8.2.2. SF-36 Statistical Analysis Method

Scores for each domain, PCS, and MCS will be summarized at each visit for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum and maximum). Differences in baseline and change from baseline between E/C/F/TAF and ABC/3TC+3rd Agent at each study visit (through Week 24) for each domain, PCS, and MCS will be assessed using a 2-sided Wilcoxon rank-sum test.

A by-subject listing for the scores for each domain, PCS, and MCS will be provided by subject ID number and visits in chronological order.

#### 8.3. HIV Treatment Satisfaction Questionnaire

The HIV Treatment Satisfaction Questionnaire (HIVTSQ) has 10 questions regarding current treatment regimen. The Status form HIVTSQs is used at Baseline, and the change form HIVTSQc is used at postbaseline visits.

#### 8.3.1. Scoring the HIV Treatment Satisfaction Questionnaire

At Baseline, a treatment satisfaction scale total will be calculated as the sum of the responses to the 10 question items on the HIVTSQs form (range from 0 to 60). At postbaseline visits, a treatment satisfaction scale total in change will be calculated as the sum of the responses to the 10 question items on the HIVTSQc form (range from -30 to 30).

Additionally, two subscale scores, one for general satisfaction/clinical and another for lifestyle/ease will be computed. Each subscale ranges from 0 to 30 on the HIVTSQs form and from -15 to 15 on the HIVTSQc form.

Table 8-1 lists the questions, possible responses for both the status and change questionnaires, as well as the subscale each question belongs to.

Table 8-1. List of Items on the HIVTSQ

| Question | Response Options for<br>Status Form | Response Options for<br>Change Form | Subscale |
|---|---|---|---|
| How satisfied are you with your current treatment? | Very satisfied 6 to 0 very dissatisfied | Much more satisfied now 3 to -3 much less satisfied now | General<br>Satisfaction/Clinical |
| How well controlled do you feel your HIV has been recently? | Very well controlled 6 to 0 very poorly controlled | Much better controlled now 3 to -3 much worse controlled now | General<br>Satisfaction/Clinical |
| How satisfied are you with any side effects of your present treatment? | Very satisfied 6 to 0 very dissatisfied | Much more satisfied now 3 to -3 much less satisfied now | General<br>Satisfaction/Clinical |
| How satisfied are you with the demands made by your current treatment? | Very satisfied 6 to 0 very dissatisfied | Much more satisfied now 3 to -3 much less satisfied now | Lifestyle/Ease |
| How convenient have you been finding your treatment to be recently? | Very convenient 6 to 0 very inconvenient | Much more convenient now 3 to -3 much less convenient now | Lifestyle/Ease |
| How flexible have you been finding your treatment to be recently? | Very flexible 6 to 0 very inflexible | Much more flexible now 3 to -3 much less flexible now | Lifestyle/Ease |
| How satisfied are you with your understanding of your HIV? | Very satisfied 6 to 0 very dissatisfied | Much more satisfied now 3 to -3 much less satisfied now | Lifestyle/Ease |
| How satisfied are you with the extent to which the treatment fits in with your lifestyle? | Very satisfied 6 to 0 very dissatisfied | Much more satisfied now 3 to -3 much less satisfied now | Lifestyle/Ease |
| Would you recommend your present treatment to someone else with HIV? | Yes I would definitely recommend the treatment 6 to 0 No I would definitely not recommend the treatment | Much more likely to recommend the treatment now 3 to -3 much less likely to recommend the treatment now | General<br>Satisfaction/Clinical |
| How satisfied would you be to continue with your present form of treatment? | Very satisfied 6 to 0 very dissatisfied | Much more satisfied now 3 to -3 much less satisfied now | General<br>Satisfaction/Clinical |

## 8.3.2. HIV Treatment Satisfaction Questionnaire Statistical Analysis Method

The HIVTSQs scale and subscale totals at baseline and each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics (n, mean, standard deviation [SD], median, Q1, Q3, minimum, and maximum). The number and percent of subjects with responses to each question will be provided at each visit.

Comparison between E/C/F/TAF and ABC/3TC+3rd Agent in HIVTSQc scale total scores will use an ANCOVA model adjusting for HIVTSQs scale total at baseline. A similar analysis will be performed on the two subscale scores as well.

For each subscale, if more than 1 question is missing, then the subscale total or subscale total in change will be set to missing. Otherwise, the missing will be imputed by taking the average of non-missing responses from the other questions in that subscale.

For the scale total or scale total in change, if more than 5 questions are missing, then the value will be set to missing. Otherwise, the missing will be imputed by taking the average of non-missing responses from the other questions.

## 8.4. Functional Assessment of Chronic Illness Therapy – Fatigue

The Functional Assessment of Chronic Illness Therapy (FACIT) was adopted from the Functional Assessment of Cancer Therapy in 1997 as an instrument to measure the health related quality of life (HRQOL) of patients with chronic illnesses. FACIT-F contains 13 additional items not in the inital FACIT questionnaire under the heading "Additional Concerns" that comprise the fatigue subscale.

The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Version 4.0 is a 40 item, self-reported questionnaire which measures the HRQOL of patients with chronic illnesses over a one-week time interval. Each item takes a range of 0 – 4, corresponding to (0) Not at all; (1) A little bit; (2) Somewhat; (3) Quite a bit; (4) Very much. Forty individual items generate 5 subscales: (1) Physical Well-Being (PWB); (2) Social/Family Well-Being (SWB); (3) Emotional Well-Being (EWB); (4) Functional Well-Being (FWB); and (5) Fatigue Subscale (FS).

### 8.4.1. Scoring the Functional Assessment of Chronic Illness Therapy – Fatigue

Full details of the scoring of the FACIT-F are available in the initial publication. A brief overview appears below. Instructions for scoring each subscale are presented in the table below. If "Reverse item?" is "Yes", then the response should be reversed by subtracting the response from "4" (ie, New response = 4 - original response).

Missing values will not be imputed. Prorating subscale scores is acceptable as long as more than 50% of items were answered (a minimum of 4 out of 7 items, 4 of 6 items, and 7 out of 13 items). This is done by multiplying the sum of the subscale by the number of items in the subscale, then dividing by the number of items actually answered.

Table 8-2. Items by Subscale and Scoring Algorithm for FACIT-F

| Subscale | Item Code | Reverse item? | Scoring Algorithm |
|---|---|---|---|
| PWB | GP1 | Yes | Sum individual item score → |
| | GP2 | Yes | Multiply by 7 → |
| | GP3 | Yes | Divide by the number of answered items (Score range: 0 - 28) |
| | GP4 | Yes | (Score range. 0 - 28) |
| | GP5 | Yes | |
| | GP6 | Yes | |
| | GP7 | Yes | |
| SWB | GS1 | No | Sum individual item score → |
| | GS2 | No | Multiply by 7 → |
| | GS3 | No | Divide by the number of answered items (Score range: 0 - 28) |
| | GS4 | No | (Score range. 0 - 20) |
| | GS5 | No | |
| | GS6 | No | |
| | GS7 | No | |
| EWB | GE1 | Yes | Sum individual item score → |
| | GE2 | No | Multiply by 6 → |
| | GE3 | Yes | Divide by the number of answered items (Score range: 0 - 24) |
| | GE4 | Yes | (Score range. 0 - 24) |
| | GE5 | Yes | |
| | GE6 | Yes | |
| FWB | GF1 | No | Sum individual item score → |
| | GF2 | No | Multiply by $7 \rightarrow$ |
| | GF3 | No | Divide by the number of answered items (Score range: 0 - 28) |
| | GF4 | No | (Score range: 0 - 20) |
| | GF5 | No | |
| | GF6 | No | |
| | GF7 | No | |
| FS | HI7 | Yes | Sum individual item score → |
| | HI12 | Yes | Multiply by 13 → |
| | An1 | Yes | Divide by the number of answered items (Score range: 0 - 52) |
| | An2 | Yes | (Score range: 0 = 32) |
| | An3 | Yes | |
| | An4 | Yes | |
| | An5 | No | |
| | An7 | No | |
| | An8 | Yes | |
| | An12 | Yes | |
| | An14 | Yes | |
| | An15 | Yes | |
| | An16 | Yes | |

Three aggregate scores can be computed as shown Table 8-3, subject to the requirements listed:

| Table 8-3. | <b>Computation of Aggregate Scores</b> |
|------------|----------------------------------------|

| Aggregate Score | Formula | Requirement |
|---|---|---|
| FACIT-F Trial Outcome Index (TOI) | PWB+FWB+FS | PWB, FWB, FS all nonmissing |
| FACT-G total score | PWB + SWB + EWB + FWB | At least 80% nonmissing (ie, 22 out of 27) |
| FACIT-F total score | PWB + SWB + EWB + FWB + FS | At least 80% nonmissing (ie, 33 out of 40) |

# 8.4.2. Functional Assessment of Chronic Illness Therapy – Fatigue Analysis Method

Scores for each subscale and aggregate score at each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum and maximum). Differences in baseline and change from baseline between E/C/F/TAF and ABC/3TC+3rd Agent for each subscale and aggregate score will be assessed at each study visit (through Week 24) using a 2-sided Wilcoxon rank-sum test.

A by-subject listing for the scores for each subscale and aggregate score will be provided by subject ID number and visits in chronological order.

#### 8.5. EQ-5D-3L

The EQ-5D-3L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale from 0 ("Worst imaginable health state") to 100 ("Best imaginable health state"). This information can be used as a quantitative measure of health outcomes as judged by the individual respondents {Rabin 2011}.

#### 8.5.1. Scoring the EQ-5D-3L Descriptive System

The scores of EQ-5D-3L descriptive system are described in the following Table 8-4.

Table 8-4. Scores of EQ-5D-3L Descriptive System

| Original Response Category | Score |
|----------------------------|-------|
| No problems | 1 |
| Some problems | 2 |
| Extreme problems | 3 |

Note: Missing values are coded as 9. Ambiguous values (eg, 2 boxes are ticked for a single dimension) should be treated as missing values.

## 8.5.2. EQ-5D Single Summary Index

EQ-5D health states, defined by the EQ-5D descriptive system, will be converted into a single summary index using the UK time trade-off (TTO) value set (Appendix 5). For example, the health state is 11111 if the response to each of the 5 dimensions of the EQ-5D system is 1. Since there are 3 possible responses (ie, 1, 2 and 3) to each of the 5 dimensions of the EQ-5D system, there are  $3^5 = 243$  health states in total.

For the UK TTO value set, the index is calculated for each of the health states (see Appendix 5 for details). Missing responses for EQ-5D-3L Questionnaire will not be imputed. If any one of the 5 dimensions is missing, the index will be missing.

## 8.5.3. Scoring the EQ VAS

For EQ VAS, the value is scored from 0 ("Worst imaginable health state") to 100 ("Best imaginable health state"). Missing values are coded as "999". Ambiguous values (eg. the line crosses the VAS twice) should be treated as missing values.

## 8.5.4. EQ-5D Statistical Analysis Method

For the 5 descriptive scores, the number and percentage of subjects with a response of "No problems", "Some problems" and "Extreme problems" will be summarized by treatment group and by baseline result for each visit. No inferential statistics will be provided.

For the index score and VAS score, change from baseline at each visit will be summarized for E/C/F/TAF, ABC/3TC+3rd Agent, and delayed switch to E/C/F/TAF. Differences in baseline and change from baseline between E/C/F/TAF and ABC/3TC+3rd Agent for the index score and VAS score will be assessed at each study visit (through Week 24) using a 2-sided Wilcoxon rank-sum test.

In addition, responder analysis will be performed based on the index score to determine the proportion of patients with health worsening or improvement by visit. Worsening or improvement in health, as measured by the proportion of patients experiencing a decrease or an increase of  $\geq 0.07$ , which is the minimally important difference (MID) {Walters 2005}, in the index score. The distribution difference in these categories between E/C/F/TAF and ABC/3TC+3rd Agent will be compared using CMH test (row mean scores differ statistic).

 Table 8-5.
 Response Category for Responder Analysis

| Response Category | Change from Baseline in Index Score |
|-------------------|-------------------------------------|
| Worsening | ≤ -0.07 |
| No change | > -0.07 and < 0.07 |
| Improvement | ≥ 0.07 |

## 9. REFERENCES

- Chan IS, Zhang Z. Test-based exact confidence intervals for the difference of two binomial proportions. Biometrics 1999;55 (4):1202-9.
- LaVange LM, Koch GG. Randomization-Based Nonparametric (ANCOVA). In: D'Agostino Sr. RB, Sullivan LM, Massaro JM, eds. Wiley Encyclopedia of Clinical Trials. John Wiley & Sons, Inc.; 2008: 31-8. vol 4).
- Maruish ME. User's manual for the SF-36v2 Health Survey. 3rd ed. Lincoln, RI: Quality Metric Incorporated.; 2011.
- Rabin R, Oemar M, Oppe M. EQ-5D-3L User Guide: Basic information on how to use the EQ-5D-3L instrument Version 4.0. EuroQol Group, 2011:
- U. S. Department of Health and Human Services, Food and Drug Administration (FDA), Center for Drug Evaluation and Research (CDER). Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment. Guidance for Industry. Silver Spring, MD. November, 2015.
- Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. Qual Life Res 2005;14 (6):1523-32.

# 10. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

nQuery Advisor(R) Version 7.0. Statistical Solutions, Cork, Ireland.

# 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

# 12. APPENDICES

| Appendix 1. | Study Procedures Table |
|---|---|
| Appendix 2. | Flowchart of US FDA-Defined Snapshot Algorithm (for Switch Study Trial) |
| Appendix 3. | Fracture Events |
| Appendix 4. | Potential Cardiovascular or Cerebrovascular Events |
| Appendix 5. | UK TTO Value Set for EQ-5D-3L Questionnaire |
| Appendix 6. | Medical History |
| Appendix 7. | Programming Specification |

**Appendix 1. Study Procedures Table** 

| | | | | | | End of | Week <sup>c</sup> | | | | 30 Day | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedure | Scrn <sup>a</sup> | Day 1 <sup>b</sup> | 4 | 8 | 12 | 24 <sup>w</sup> | 28 <sup>d</sup> | 32 <sup>d</sup> | 36 | 48 | Follow-up <sup>e</sup> | ESDD <sup>f</sup> |
| Informed Consent | X | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X |
| Complete Physical Exam <sup>g</sup> | X | X | | | | X | | | | X | | X |
| Symptom-Directed Physical Exam <sup>h</sup> | | | X | X | X | | X | X | X | | X | |
| 12-Lead ECG (Performed Supine) | X | | | | | | | | | X | | X |
| Vital Signs and Weight | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | |
| Urinalysis and Urine Chemistry | X | X | X | X | X | X | X | X | X | X | X <sup>u</sup> | X |
| Urine Storage Sample | | X | X | X | X | X | X | X | X | X | | X |
| Urine Pregnancy Test <sup>i</sup> | | X | X | X | X | X | X | X | X | X | X | X |
| Serum Pregnancy Test <sup>i</sup> | X | | | | | | | | | | | |
| Chemistry Profile <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology Profile <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| Plasma HIV-1 RNA <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| CD4+ Cell Count | X | X | X | X | X | X | X | X | X | X | X | X |
| Whole Blood Sample <sup>m</sup> | X | | | | | | | | | | | |
| HBV and HCV Serologies <sup>n</sup> | X | | | | | | | | | | | |
| Metabolic Assessments <sup>o</sup> | | X | | X | X | | | | $X^d$ | X | | |
| Cystatin C | | X | | | | | | | | | | |

| | | | | | | End of | Week | | | | 30 Day | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedure | Scrna | Day 1 <sup>b</sup> | 4 | 8 | 12 | 24 <sup>w</sup> | 28 <sup>d</sup> | 32 <sup>d</sup> | 36 | 48 | Follow-up <sup>e</sup> | ESDD <sup>f</sup> |
| Estimated GFR <sub>CG</sub> <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | | X |
| Plasma Sample Storageq | | X | X | X | X | X | X | X | X | X | | X |
| PPD | | X | X | | X | X | X | | X <sup>d</sup> | X | | X |
| HIV-1 Genotype/Phenotyper | | | | | | | | | | X | | X |
| Evaluations of Bone & Renal Safety, Inflammation and Platelet and Coagulation Functions | | X | X | | X | X | X | | $X^d$ | X | | X |
| Questionnaires: VAS, HIVTSQs, HIVTSQc, EQ-5D, SF-36, and FACIT-F <sup>t</sup> | | X | X | X | X | X | X | X | X | X | | X |
| Randomization | | X | | | | | | | | | | |
| Study Drug Dispensation and Accountability | | X | X | X | X | X | X | | X <sup>v</sup> | | | X <sup>v</sup> |

- a Evaluations to be completed within 42 days prior to the Day 1 visit
- b Subjects will be dispensed study drug on the Day 1 visit; initiation of treatment with the study drug must take place within 24h ours after the Day 1 visit. E/C/F/TAF FDC will be provided to subjects randomized to Treatment Group 1.
- c All study visits are to be scheduled relative to the Day 1 visit date. Visit windows are  $\pm$  2 days of the protocol specified date through Week 12,  $\pm$  6 days of the protocol specified date. Unless notified by Gilead, the Week 48 visit should be completed within  $\pm$  6 days of the visit date. For Treatment Group 2 subjects, the Weeks 28 and 32 visit windows are  $\pm$  2 days of the protocol specified date.
- d Treatment Group 2 subjects only
- e Only required for those subjects who permanently discontinue study drug or their current regimen and refuse continue study visits through Week 48. For the purpose of scheduling a 30-Day Follow-Up Visit, a ± 6 days window may be used.
- f Early Study Drug Discontinuation visit to occur within 72 hours of last dose of study drug. Subjects will be asked to continue attending the scheduled study visits through Week 48 visit even if the subject discontinues study drug.
- g Complete physical examination (urogenital/anorectal exams will be performed at the discretion of the Investigator)
- h Symptom-directed physical examination as needed
- i Females of childbearing potential only. Positive urine pregnancy tests will be confirmed with a serum test.
- j Chemistry profile: alkaline phosphatase, AST, ALT, total bilirubin, direct and indirect bilirubin, total protein, albumin, bicarbonate, BUN, calcium, chloride, creatinine, glucose, potassium, and sodium. At visits in which metabolic assessments are to be performed, analyses of glucose will be done as part of the fasting metabolic assessments and not as part of the chemistry profile.
- k CBC with differential and platelet count
- If the HIV-1 RNA value is ≥ 50 copies/mL, a retest should be collected at a scheduled or unscheduled visit, 2-4 weeks after the date of the original test (except for screening and Day 1 results). HIV-1 genotype/phenotype resistance testing only conducted for subjects with confirmed virologic failure with HIV-1 RNA value ≥ 50 copies/mL. Subjects should be managed according to Figure 6-1 in the protocol.

- m Whole blood sample for proviral genotype analysis of archived resistance (if historical plasma genotype report prior to first ARV is not available or subject has 3 or more ART regimens)
- n Hepatitis B virus surface Antigen (HBsAg), Hepatitis B core antibody (HBcAb), and Hepatitis C virus (HCV Ab) serologies (reflex HCV RNA is performed in subjects with positive HCVAb serology)
- o Metabolic Assessments: Metabolic Assessments: Fasting glucose and lipid panel (total cholesterol, HDL, direct LDL, triglycerides). If the subject has not fasted prior to the visit, the visit may proceed, but the subject must return within 72 hours in a fasted state.
- p Estimated GFR according to the Cockcroft-Gault formula for creatinine clearance
- q PPD
- r HIV-1 genotype/phenotype resistance testing for subjects with unconfirmed virologic rebound with HIV-1 RNA value ≥ 50 copies/mL
- s Blood for bone safety, parathyroid hormone (PTH) and serum OH-25 vitamin D. Urine for renal safety, including retinol binding protein, and beta-2-microglobulin, will be collected. Samples will be collected fasted. If the subject has not fasted prior to the visit, the visit may proceed, but the subject must return within 72 hours in a fasted state.
- t EQ-5D, SF-36, and FACIT F will be administered at Day 1, Weeks 4, 24, 28 (Treatment Group 2 only) and 48. HIVTSQs will be administered on Day 1. HIVTSQc will be administered at Weeks 4, 12, 24, 28 (Treatment Group 2 only) 48 and ESDD. VAS will be administered at the following visits: Day 1 Week 48 and ESDD.
- u Urinalysis only
- v Drug accountability only; study drug will not be dispensed at this visit.
- w At Week 24, subjects randomized to Treatment Group 2 will discontinue their current regimen of ABC/3TC plus a third antiretroviral agent and will switch to E/C/F/TAF FDC; initiation of treatment with the study drug must take place within 24 hours after the Week 24 visit. E/C/F/TAF FDC will be provided to subjects.

# Appendix 2. Flowchart of US FDA-Defined Snapshot Algorithm (for Switch Study Trial)

The following flowchart for US FDA-defined snapshot algorithm is based on the US FDA Guidance on Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for treatment {U. S. Department of Health and Human Services 2015}



<sup>\*</sup> On-Treatment HIV-1 RNA data include all HIV-1 RNA data for subjects who are on-going and HIV-1 RNA data up to 1 day after the last dose date of study drug for subjects who prematurely discontinue or complete study drug.

## **Appendix 3.** Fracture Events

The selected PTs from SMQ of Osteoporosis/Osteopenia and HLGT of fractures based on clinical review are listed as follows.

| | Selected PTs Based on SMQ of Osteoporosis/Osteopenia | Selected PTs Based on HLGT of Fractures |
|---|---|---|
| 1 | Acetabulum Fracture | Acetabulum fracture |
| 2 | Atypical Femur Fracture | Atypical femur fracture |
| 3 | Cervical Vertebral Fracture | Cervical vertebral fracture |
| 4 | Femoral Neck Fracture | Femoral neck fracture |
| 5 | Femur Fracture | Femur fracture |
| 6 | Forearm Fracture | Forearm fracture |
| 7 | Fracture | Fracture |
| 8 | Fractured Ischium | Fractured ischium |
| 9 | Fractured Sacrum | Fractured sacrum |
| 10 | Hip Fracture | Hip fracture |
| 11 | Ilium Fracture | Ilium fracture |
| 12 | Lumbar Vertebral Fracture | Lumbar vertebral fracture |
| 13 | Multiple Fractures | Multiple fractures |
| 14 | Osteoporotic Fracture | Osteoporotic fracture |
| 15 | Pathological Fracture | Pathological fracture |
| 16 | Pelvic Fracture | Pelvic fracture |
| 17 | Pubis Fracture | Pubis fracture |
| 18 | Radius Fracture | Radius fracture |
| 19 | Rib Fracture | Rib fracture |
| 20 | Sacroiliac Fracture | Sacroiliac fracture |
| 21 | Spinal Compression Fracture | Spinal compression fracture |
| 22 | Spinal Fracture | Spinal fracture |
| 23 | Thoracic Vertebral Fracture | Thoracic vertebral fracture |
| 24 | Wrist Fracture | Wrist fracture |
| 25 | Closed Fracture Manipulation | Ankle fracture |
| 26 | External Fixation of Fracture | Atypical fracture |
| 27 | Fracture Treatment | Avulsion fracture |
| 28 | Internal Fixation of Fracture | Bone fissure |
| 29 | Open Reduction of Fracture | Bone fragmentation |
| 30 | Open Reduction of Spinal Fracture | Chance fracture |
| 31 | Tartrate-resistant acid phosphatase decreased | Clavicle fracture |
| 32 | Vertebral Body Replacement | Comminuted fracture |
| 33 | Vertebroplasty | Complicated fracture |

| | Selected PTs Based on SMQ of Osteoporosis/Osteopenia | Selected PTs Based on HLGT of Fractures |
|---|---|---|
| 34 | | Compression fracture |
| 35 | | Craniofacial fracture |
| 36 | | Epiphyseal fracture |
| 37 | | Facial bones fracture |
| 38 | | Fibula fracture |
| 39 | | Flail chest |
| 40 | | Foot fracture |
| 41 | | Fracture displacement |
| 42 | | Fracture of clavicle due to birth trauma |
| 43 | | Fractured coccyx |
| 44 | | Fractured skull depressed |
| 45 | | Greenstick fracture |
| 46 | | Hand fracture |
| 47 | | Humerus fracture |
| 48 | | Impacted fracture |
| 49 | | Jaw fracture |
| 50 | | Limb fracture |
| 51 | | Lower limb fracture |
| 52 | | Open fracture |
| 53 | | Osteochondral fracture |
| 54 | | Patella fracture |
| 55 | | Periprosthetic fracture |
| 56 | | Scapula fracture |
| 57 | | Scapulothoracic dissociation |
| 58 | | Skull fracture |
| 59 | | Skull fractured base |
| 60 | | Sternal fracture |
| 61 | | Stress fracture |
| 62 | | Tibia fracture |
| 63 | | Torus fracture |
| 64 | | Traumatic fracture |
| 65 | | Ulna fracture |
| 66 | | Upper limb fracture |

Note: AEs are coded by MedDRA 20.1.

## **Appendix 4.** Potential Cardiovascular or Cerebrovascular Events

The selected PTs of potential cardiovascular or cerebrovascular events based on clinical review are listed as follows.

| | Selected PTs Based on Clinical Review | | Selected PTs Based on Clinical Review |
|---|---|---|---|
| 1 | Acute coronary syndrome | 93 | Coronary endarterectomy |
| 2 | Acute myocardial infarction | 94 | Coronary no-reflow phenomenon |
| 3 | Amaurosis fugax | 95 | Coronary ostial stenosis |
| 4 | Angina pectoris | 96 | Coronary revascularisation |
| 5 | Angina unstable | 97 | Coronary vascular graft occlusion |
| 6 | Anginal equivalent | 98 | Coronary vascular graft stenosis |
| 7 | Arteriogram coronary abnormal | 99 | Delayed ischaemic neurological deficit |
| 8 | Arteriosclerosis coronary artery | 100 | Dissecting coronary artery aneurysm |
| 9 | Arteriospasm coronary | 101 | ECG electrically inactive area |
| 10 | Basal ganglia infarction | 102 | ECG signs of myocardial infarction |
| 11 | Basal ganglia stroke | 103 | ECG signs of myocardial ischaemia |
| 12 | Basilar artery occlusion | 104 | Electrocardiogram Q wave abnormal |
| 13 | Basilar artery stenosis | 105 | Electrocardiogram ST segment abnormal |
| 14 | Basilar artery thrombosis | 106 | Electrocardiogram ST segment depression |
| 15 | Blood creatine phosphokinase abnormal | 107 | Electrocardiogram ST segment elevation |
| 16 | Blood creatine phosphokinase increased | 108 | Electrocardiogram ST-T segment abnormal |
| 17 | Blood creatine phosphokinase MB abnormal | 109 | Electrocardiogram ST-T segment depression |
| 18 | Blood creatine phosphokinase MB increased | 110 | Electrocardiogram ST-T segment elevation |
| 19 | Brachiocephalic arteriosclerosis | 111 | Electrocardiogram T wave abnormal |
| 20 | Brachiocephalic artery occlusion | 112 | Electrocardiogram T wave inversion |
| 21 | Brachiocephalic artery stenosis | 113 | Electrocardiogram U wave inversion |
| 22 | Brain hypoxia | 114 | Embolic cerebral infarction |
| 23 | Brain stem embolism | 115 | Embolic stroke |
| 24 | Brain stem infarction | 116 | Exercise electrocardiogram abnormal |
| 25 | Brain stem ischaemia | 117 | Exercise test abnormal |
| 26 | Brain stem stroke | 118 | External counterpulsation |
| 27 | Brain stem thrombosis | 119 | Haemorrhage coronary artery |
| 28 | Capsular warning syndrome | 120 | Hypoxic-ischaemic encephalopathy |
| 29 | Cardiac stress test abnormal | 121 | Infarction |

| | Selected PTs Based on Clinical Review | | Selected PTs Based on Clinical Review |
|---|---|---|---|
| 30 | Cardiac ventricular scarring | 122 | Inner ear infarction |
| 31 | Cardiopulmonary exercise test abnormal | 123 | Ischaemic cardiomyopathy |
| 32 | Carotid angioplasty | 124 | Ischaemic cerebral infarction |
| 33 | Carotid arterial embolus | 125 | Ischaemic mitral regurgitation |
| 34 | Carotid arteriosclerosis | 126 | Ischaemic stroke |
| 35 | Carotid artery bypass | 127 | Kounis syndrome |
| 36 | Carotid artery calcification | 128 | Lacunar infarction |
| 37 | Carotid artery disease | 129 | Lacunar stroke |
| 38 | Carotid artery insufficiency | 130 | Lateral medullary syndrome |
| 39 | Carotid artery occlusion | 131 | Microvascular coronary artery disease |
| 40 | Carotid artery restenosis | 132 | Migrainous infarction |
| 41 | Carotid artery stenosis | 133 | Millard-Gubler syndrome |
| 42 | Carotid artery stent insertion | 134 | Moyamoya disease |
| 43 | Carotid artery stent removal | 135 | Myocardial hypoxia |
| 44 | Carotid artery thrombosis | 136 | Myocardial infarction |
| 45 | Carotid endarterectomy | 137 | Myocardial ischaemia |
| 46 | Carotid revascularisation | 138 | Myocardial necrosis |
| 47 | Cerebellar artery occlusion | 139 | Myocardial necrosis marker increased |
| 48 | Cerebellar artery thrombosis | 140 | Myocardial reperfusion injury |
| 49 | Cerebellar embolism | 141 | Myocardial stunning |
| 50 | Cerebellar infarction | 142 | Papillary muscle infarction |
| 51 | Cerebellar ischaemia | 143 | Percutaneous coronary intervention |
| 52 | Cerebellar stroke | 144 | Perinatal stroke |
| 53 | Cerebral arteriosclerosis | 145 | Periprocedural myocardial infarction |
| 54 | Cerebral artery embolism | 146 | Post angioplasty restenosis |
| 55 | Cerebral artery occlusion | 147 | Post cardiac arrest syndrome |
| 56 | Cerebral artery restenosis | 148 | Post procedural myocardial infarction |
| 57 | Cerebral artery stenosis | 149 | Post procedural stroke |
| 58 | Cerebral artery thrombosis | 150 | Postinfarction angina |
| 59 | Cerebral gas embolism | 151 | Precerebral arteriosclerosis |
| 60 | Cerebral infarction | 152 | Precerebral artery occlusion |
| 61 | Cerebral infarction foetal | 153 | Prinzmetal angina |
| 62 | Cerebral ischaemia | 154 | Reversible cerebral vasoconstriction syndrome |

| | Selected PTs Based on Clinical Review | | Selected PTs Based on Clinical Review |
|---|---|---|---|
| 63 | Cerebral microembolism | 155 | Reversible ischaemic neurological deficit |
| 64 | Cerebral revascularisation | 156 | Scan myocardial perfusion abnormal |
| 65 | Cerebral septic infarct | 157 | Silent myocardial infarction |
| 66 | Cerebral small vessel ischaemic disease | 158 | Spinal artery embolism |
| 67 | Cerebral thrombosis | 159 | Spinal artery thrombosis |
| 68 | Cerebral vascular occlusion | 160 | Stress cardiomyopathy |
| 69 | Cerebral vasoconstriction | 161 | Stress echocardiogram abnormal |
| 70 | Cerebral venous thrombosis | 162 | Stroke in evolution |
| 71 | Cerebrovascular accident | 163 | Subclavian coronary steal syndrome |
| 72 | Cerebrovascular disorder | 164 | Subclavian steal syndrome |
| 73 | Cerebrovascular insufficiency | 165 | Subendocardial ischaemia |
| 74 | Cerebrovascular stenosis | 166 | Thalamic infarction |
| 75 | Computerised tomogram coronary artery abnormal | 167 | Thrombotic cerebral infarction |
| 76 | Coronary angioplasty | 168 | Thrombotic stroke |
| 77 | Coronary arterial stent insertion | 169 | Transient ischaemic attack |
| 78 | Coronary artery bypass | 170 | Troponin I increased |
| 79 | Coronary artery compression | 171 | Troponin increased |
| 80 | Coronary artery disease | 172 | Troponin T increased |
| 81 | Coronary artery dissection | 173 | Vascular encephalopathy |
| 82 | Coronary artery embolism | 174 | Vascular graft occlusion |
| 83 | Coronary artery insufficiency | 175 | Vascular stent occlusion |
| 84 | Coronary artery occlusion | 176 | Vascular stent restenosis |
| 85 | Coronary artery reocclusion | 177 | Vascular stent stenosis |
| 86 | Coronary artery restenosis | 178 | Vascular stent thrombosis |
| 87 | Coronary artery stenosis | 179 | Vertebral artery occlusion |
| 88 | Coronary artery surgery | 180 | Vertebral artery stenosis |
| 89 | Coronary artery thrombosis | 181 | Vertebral artery thrombosis |
| 90 | Coronary brachytherapy | 182 | Vertebrobasilar insufficiency |
| 91 | Coronary bypass stenosis | 183 | Wall motion score index abnormal |
| 92 | Coronary bypass thrombosis | | |

Note: AEs are coded by MedDRA 20.1.

### Appendix 5. UK TTO Value Set for EQ-5D-3L Questionnaire

For the UK TTO value set, the index is calculated for each of the health states based on the following equation:

Index = 1 - 0.081 - 0.069 MO2 - 0.314 MO3 - 0.104 SC2 - 0.214 SC3 - 0.036 UA2 - 0.094 UA3 - 0.123 PD2 - 0.386 PD3 - 0.071 AD2 - 0.236 AD3 - 0.269 N3

- -0.081 is a constant term for any dysfunctional state.
- MO2 is a dummy variable for level 2 of Mobility.
- MO3 is a dummy variable for level 3 of Mobility.
- SC2 is a dummy variable for level 2 of Self Care.
- SC3 is a dummy variable for level 3 of Self Care.
- UA2 is a dummy variable for level 2 of Usual Activities.
- UA3 is a dummy variable for level 3 of Usual Activities.
- PD2 is a dummy variable for level 2 of Pain/Discomfort.
- PD3 is a dummy variable for level 3 of Pain/Discomfort.
- AD2 is a dummy variable for level 2 of Anxiety/Depression.
- AD3 is a dummy variable for level 3 of Anxiety/Depression.
- N3 is a dummy variable that represents level 3 occurs within at least one dimension.

The index score is missing if any one of the 5 dimensions is missing.

| UK TTO | | | | | |
|---|---|---|---|---|---|
| <b>Health State</b> | <b>Index Value</b> | Health State | <b>Index Value</b> | Health State | Index Value |
| 11111 | 1.000 | 12233 | -0.112 | 21132 | 0.124 |
| 11112 | 0.848 | 12311 | 0.452 | 21133 | -0.041 |
| 11113 | 0.414 | 12312 | 0.381 | 21211 | 0.814 |
| 11121 | 0.796 | 12313 | 0.216 | 21212 | 0.743 |
| 11122 | 0.725 | 12321 | 0.329 | 21213 | 0.309 |
| 11123 | 0.291 | 12322 | 0.258 | 21221 | 0.691 |
| 11131 | 0.264 | 12323 | 0.093 | 21222 | 0.620 |
| 11132 | 0.193 | 12331 | 0.066 | 21223 | 0.186 |
| 11133 | 0.028 | 12332 | -0.005 | 21231 | 0.159 |
| 11211 | 0.883 | 12333 | -0.170 | 21232 | 0.088 |
| 11212 | 0.812 | 13111 | 0.436 | 21233 | -0.077 |
| 11213 | 0.378 | 13112 | 0.365 | 21311 | 0.487 |
| 11221 | 0.760 | 13113 | 0.200 | 21312 | 0.416 |
| 11222 | 0.689 | 13121 | 0.313 | 21313 | 0.251 |
| 11223 | 0.255 | 13122 | 0.242 | 21321 | 0.364 |
| 11231 | 0.228 | 13123 | 0.077 | 21322 | 0.293 |
| 11232 | 0.157 | 13131 | 0.050 | 21323 | 0.128 |
| 11233 | -0.008 | 13132 | -0.021 | 21331 | 0.101 |
| 11311 | 0.556 | 13133 | -0.186 | 21332 | 0.030 |
| 11312 | 0.485 | 13211 | 0.400 | 21333 | -0.135 |
| 11313 | 0.320 | 13212 | 0.329 | 22111 | 0.746 |
| 11321 | 0.433 | 13213 | 0.164 | 22112 | 0.675 |
| 11322 | 0.362 | 13221 | 0.277 | 22113 | 0.241 |
| 11323 | 0.197 | 13222 | 0.206 | 22121 | 0.623 |
| 11331 | 0.170 | 13223 | 0.041 | 22122 | 0.552 |
| 11332 | 0.099 | 13231 | 0.014 | 22123 | 0.118 |
| 11333 | -0.066 | 13232 | -0.057 | 22131 | 0.091 |
| 12111 | 0.815 | 13233 | -0.222 | 22132 | 0.020 |
| 12112 | 0.744 | 13311 | 0.342 | 22133 | -0.145 |
| 12113 | 0.310 | 13312 | 0.271 | 22211 | 0.710 |
| 12121 | 0.692 | 13313 | 0.106 | 22212 | 0.639 |
| 12122 | 0.621 | 13321 | 0.219 | 22213 | 0.205 |
| 12123 | 0.187 | 13322 | 0.148 | 22221 | 0.587 |
| 12131 | 0.160 | 13323 | -0.017 | 22222 | 0.516 |
| 12132 | 0.089 | 13331 | -0.044 | 22223 | 0.082 |
| 12133 | -0.076 | 13332 | -0.115 | 22231 | 0.055 |
| 12211 | 0.779 | 13333 | -0.280 | 22232 | -0.016 |
| 12212 | 0.708 | 21111 | 0.850 | 22233 | -0.181 |
| 12213 | 0.274 | 21112 | 0.779 | 22311 | 0.383 |
| 12221 | 0.656 | 21113 | 0.345 | 22312 | 0.312 |
| 12222 | 0.585 | 21121 | 0.727 | 22313 | 0.147 |
| 12223 | 0.151 | 21122 | 0.656 | 22321 | 0.260 |
| 12231 | 0.124 | 21123 | 0.222 | 22322 | 0.189 |
| 12232 | 0.053 | 21131 | 0.195 | 22323 | 0.024 |

| UK TTO | | | | | |
|---|---|---|---|---|---|
| <b>Health State</b> | <b>Index Value</b> | Health State | <b>Index Value</b> | Health State | Index Value |
| 22331 | -0.003 | 31223 | -0.059 | 33122 | -0.072 |
| 22332 | -0.074 | 31231 | -0.086 | 33123 | -0.237 |
| 22333 | -0.239 | 31232 | -0.157 | 33131 | -0.264 |
| 23111 | 0.367 | 31233 | -0.322 | 33132 | -0.335 |
| 23112 | 0.296 | 31311 | 0.242 | 33133 | -0.500 |
| 23113 | 0.131 | 31312 | 0.171 | 33211 | 0.086 |
| 23121 | 0.244 | 31313 | 0.006 | 33212 | 0.015 |
| 23122 | 0.173 | 31321 | 0.119 | 33213 | -0.150 |
| 23123 | 0.008 | 31322 | 0.048 | 33221 | -0.037 |
| 23131 | -0.019 | 31323 | -0.117 | 33222 | -0.108 |
| 23132 | -0.090 | 31331 | -0.144 | 33223 | -0.273 |
| 23133 | -0.255 | 31332 | -0.215 | 33231 | -0.300 |
| 23211 | 0.331 | 31333 | -0.380 | 33232 | -0.371 |
| 23212 | 0.260 | 32111 | 0.232 | 33233 | -0.536 |
| 23213 | 0.095 | 32112 | 0.161 | 33311 | 0.028 |
| 23221 | 0.208 | 32113 | -0.004 | 33312 | -0.043 |
| 23222 | 0.137 | 32121 | 0.109 | 33313 | -0.208 |
| 23223 | -0.028 | 32122 | 0.038 | 33321 | -0.095 |
| 23231 | -0.055 | 32123 | -0.127 | 33322 | -0.166 |
| 23232 | -0.126 | 32131 | -0.154 | 33323 | -0.331 |
| 23233 | -0.291 | 32132 | -0.225 | 33331 | -0.358 |
| 23311 | 0.273 | 32133 | -0.390 | 33332 | -0.429 |
| 23312 | 0.202 | 32211 | 0.196 | 33333 | -0.594 |
| 23313 | 0.037 | 32212 | 0.125 | | |
| 23321 | 0.150 | 32213 | -0.040 | | |
| 23322 | 0.079 | 32221 | 0.073 | | |
| 23323 | -0.086 | 32222 | 0.002 | | |
| 23331 | -0.113 | 32223 | -0.163 | | |
| 23332 | -0.184 | 32231 | -0.190 | | |
| 23333 | -0.349 | 32232 | -0.261 | | |
| 31111 | 0.336 | 32233 | -0.426 | | |
| 31112 | 0.265 | 32311 | 0.138 | | |
| 31113 | 0.100 | 32312 | 0.067 | | |
| 31121 | 0.213 | 32313 | -0.098 | | |
| 31122 | 0.142 | 32321 | 0.015 | | |
| 31123 | -0.023 | 32322 | -0.056 | | |
| 31131 | -0.050 | 32323 | -0.221 | | |
| 31132 | -0.121 | 32331 | -0.248 | | |
| 31133 | -0.286 | 32332 | -0.319 | | |
| 31211 | 0.300 | 32333 | -0.484 | | |
| 31212 | 0.229 | 33111 | 0.122 | | |
| 31213 | 0.064 | 33112 | 0.051 | | |
| 31221 | 0.177 | 33113 | -0.114 | | |
| 31222 | 0.106 | 33121 | -0.001 | | |

### **Appendix 6.** Medical History

The following medical history will be summarized.

- **Diabetes Mellitus (Yes/No):** "Yes" includes subjects with at least one of the following medical condition terms: diabetes, diabetes mellitus, diabetes 1, diabetes 2, Type 1 Diabetes, Type 2 Diabetes.
- **Hypertension (Yes/No):** "Yes" includes subjects with at least one of the following medical conditions: hypertension, blood pressure, high blood pressure, elevated blood pressure.
- Cardiovascular Disease (Yes/No): "Yes" includes subjects with at least one of the following medical conditions: cardiovascular disease, coronary artery disease, myocardial infarction, angina, cardiac ischemia, transient ischemic attack, stroke, claudication, peripheral vascular disease.
- **Hyperlipidemia (Yes/No):** "Yes" includes subjects with at least one of the following medical conditions: hyperlipidemia, lipids elevated, hypercholesterolemia, cholesterol elevated, LDL elevated, hypertriglyceridemia, triglycerides elevated.

The selected medical condition terms from the MH dataset or preferred terms from the AE dataset for a subject having the medical risk factors of interest are listed as follows:

| | Medical Conditions from MH Dataset | | | |
|---|---|---|---|---|
| | Hypertension | Diabetes | Cardiovascular Disease | Hyperlipidemia |
| 1 | ARTERIAL<br>HYPERTENSION | ADULT ONSET<br>DIABETES MELLITUS | ACUTE MYOCARDIAL INFARCTION | CHRONIC<br>HYPERCHOLESTEROLE<br>MIA |
| 2 | BENIGN ESSENTIAL<br>HYPERTENSION | ADULT ONSET<br>DIABETES MELLITUS<br>(TYPE 2) | ANGINA | DIABETES MELLITUS<br>TYPE I WITH<br>HYPERLIPIDEMIA |
| 3 | BENIGN<br>HYPERTENSION | BORDERLINE DIABETES<br>MELLITUS TYPE II | CORONARY ARTERY<br>BYPASS GRAFT | DYSLIPIDEMAIA |
| 4 | BORDERLINE<br>HYPERTENSION | DIABETES | CORONARY ARTERY<br>DISEASE | DYSLIPIDEMIA |
| 5 | ELEVATED BLOOD<br>PRESSURE | DIABETES INSULIN<br>DEPENDENT | CORONARY DISEASE | DYSLIPIDEMIE |
| 6 | ELEVATED BLOOD<br>PRESSURE READING<br>WITHOUT DIAGNOSIS<br>OF HYPERTENSION | DIABETES - TYPE 2 | CORONARY HEART<br>DISEASE | ELEVATED<br>CHOLESTEROL |
| 7 | ELEVATED BLOOD<br>PRESSURE WITHOUT<br>DIAGNOSIS | DIABETES MELISTUS<br>TYPE II | CORONARY STENTS | ELEVATED<br>TRIGLYCERIDES |
| 8 | ELEVATED BLOOD<br>PRESSURE WITHOUT<br>DIAGNOSIS OF<br>HYPERTENSION | DIABETES MELLITIS<br>TYPE 1 | CORONARY TRIPLE<br>BYPASS | FAMILIAL HYPER-<br>CHOLESTEROLAEMIA |

| | Medical Conditions from MH Dataset | | | |
|---|---|---|---|---|
| | Hypertension | Diabetes | Cardiovascular Disease | Hyperlipidemia |
| 9 | ESSENTIAL<br>HYPERTENSION | DIABETES MELLITIS<br>TYPE II | CORONNARY ARTERY<br>DISEASE | HIGH CHOLESTEROL |
| 10 | ESSENTIAL<br>HYPERTENSION,<br>BENIGN | DIABETES MELLITUS | HYPERTENSVE<br>CARDIOPATHY | HIGH TRIGLYCERIDES |
| 11 | HIGH BLOOD PRESSURE | DIABETES MELLITUS<br>TYPE II | INFERIOR WALL<br>MYOCARDIAL<br>INFARCTION | HYLERLIPIDEMIA |
| 12 | HIGH BLOOD PRESSURE<br>(WHEN AT MD OFFICE -<br>NO DIAGNOSIS OF<br>HYPERTENSION | DIABETES MELLITUS<br>(ADULT ONSET/TYPE 2) | INTERMITTENT<br>CLAUDICATION OF THE<br>LOWER EXTREMITIES | HYPER-<br>CHOLESTERALEMIA |
| 13 | HYPER TENSION | DIABETES MELLITUS<br>(TYPE 2) | ISCHEMIC LEFT GREAT<br>TOE | HYPERCHOLESTEREMIA |
| 14 | HYPERTENSION | DIABETES MELLITUS 2 | LEFT MIDDLE<br>CEREBRAL ARTERY<br>STROKE | HYPERCHOLESTEROL |
| 15 | HYPERTENSION<br>(DIAGNOSED BY<br>COMPUTERIZED<br>MONITORING) | DIABETES MELLITUS II | MILD CORONARY<br>ATHEROSCLEROSIS | HYPER-<br>CHOLESTEROLEMIA |
| 16 | HYPERTENSION<br>(SELF REPORTED) | DIABETES MELLITUS<br>TYP II | MYOCARDIAL<br>INFARCTION | HYPER-<br>CHOLESTERONEMIA |
| 17 | HYPERTENSION<br>ARTERIAL | DIABETES MELLITUS<br>TYPE 2 | MYOCARDIAL<br>INFARCTION,PCI AND<br>STENT | HYPERLIMIDEMIA |
| 18 | HYPERTENSION IN<br>TREATMENT | DIABETES MELLITUS<br>TYPE I WITH<br>HYPERLIPIDEMIA | NON-ISCHEMIC<br>CARDIOMYOPATHY | HYPERLIPDEMIA |
| 19 | HYPERTENSION<br>RELATED TO<br>EMOTIONS | DIABETES MELLITUS<br>TYPE II | OLD MYOCARDIAL<br>INFARCTION | HYPERLIPEDEMIA |
| 20 | HYPERTENSION,<br>BENIGN ESSENTIAL | DIABETES MELLITUS<br>TYPE II, WITHOUT<br>RETINOPATHY | POSSIBLE<br>CEREBROVASCULAR<br>ACCIDENT HISTORY | HYPERLIPIDEMIA |
| 21 | HYPERTENSIVE | DIABETES MELLITUS,<br>TYPE II | POSSIBLE<br>MYOCARDIAL<br>INFARCTION HISTORY | HYPERLIPIDEMIA<br>(COMBINED) |
| 22 | HYPERTENSVE<br>CARDIOPATHY | DIABETES MILLITUS II | TRANSIENT ISCHAEMIC<br>ATTACK | HYPERLIPIMIA |
| 23 | HYPERTENTION | DIABETES TYPE 1 | TRANSIENT ISCHEMIC<br>ATTACK | HYPER-<br>CHOLESTEROLEMIA |
| 24 | INCREASED BLOOD<br>PRESSURE | DIABETES TYPE 2 | VASOSPASTIC ANGINA<br>WITH NON ST<br>ELEVATION MI | HYPERTRIGLICEREMIA |

| | Medical Conditions from MH Dataset | | | |
|---|---|---|---|---|
| | Hypertension | Diabetes | Cardiovascular Disease | Hyperlipidemia |
| 25 | INTERMITTENT<br>INCREASED BLOOD<br>PRESSURE | DIABETES TYPE II | | HYPERTRIGLYCERIDEMIA |
| 26 | INTERMKTTENT<br>INCREASED BLOOD<br>PRESSURE | DIABETES, TYPE II | | MIXED<br>HYPERLIPIDEMIA |
| 27 | ISOLATED HIGH BLOOD<br>PRESSURE EPISODE | DIABETIC COMA | | RAISED CHOLESTEROL |
| 28 | STRESS INDUCED<br>HYPERTENSION | DIABETIC ERECTILE<br>DYSFUNCTION | | |
| 29 | | DIABETIC FOOT | | |
| 30 | | DIABETIC<br>NEUROPATHIC | | |
| 31 | | DIABETIC<br>NEUROPATHY | | |
| 32 | | DIABETIC PERIPHERAL<br>NEUROPATHY | | |
| 33 | | DIABETIC<br>RETINOPATHY | | |
| 34 | | DIABETIES | | |
| 34 | | FAMILIARITY FOR<br>DIABETES MELLITUS<br>TYPE II | | |
| 36 | | FAMILY HISTORY FOR DIABETES | | |
| 37 | | GESTATIMEL DIABETES | | |
| 38 | | HYPERGLYCEMIA | | |
| 39 | | MELLITUS DIABETES IN TREATMENT | | |
| 40 | | NON INSULIN<br>DEPENDENT DIABETES<br>MELLITUS | | |
| 41 | | NONINSULIN-DEPENDENT<br>DIABETES MELLITUS | | |
| 42 | | PROTEINURIA<br>(RELATED TO DIABETES<br>PER NEPHROLOGIST<br>PER SUBJECT) | | |
| 43 | | TYPE 2 DIABETE | | |
| 44 | | TYPE 2 DIABETES | | |
| 45 | | TYPE 2 DIABETES<br>MELLITUS | | |
| 46 | | TYPE II DIABETES | | |

| | MedDRA Preferred Terms from AE Dataset | | | |
|---|---|---|---|---|
| | Hypertension | Diabetes | Cardiovascular Disease | Hyperlipidemia |
| 1 | Blood pressure inadequately controlled | Diabetes mellitus | Acute myocardial infarction | Hyperlipidemia |
| 2 | Blood pressure increased | Type 2 diabetes mellitus | Cardiac arrest | Blood cholesterol increased |
| 3 | Hypertension | | Cerebral infarction | Dyslipidaemia |
| 4 | Hypertensive crisis | | Cerebrovascular accident | Hypercholesterolaemia |
| 5 | | | Coronary artery disease | Hyperlipidaemia |
| 6 | | | Electrocardiogram abnormal | Hypertriglyceridaemia |
| 7 | | | Enlarged uvula | Lipids abnormal |
| 8 | | | Haemorrhagic transformation stroke | Type V hyperlipidaemia |
| 9 | | | Left ventricular dysfunction | |
| 10 | | | Myocardial ischaemia | |
| 11 | | | Peripheral ischaemia | |

The selected combination of medication class and indication from the CM dataset for a subject having the medical risk factors of interest are listed as follows:

| | Medication Class | Indication |
|---|---|---|
| | Нурег | tension |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ANTIHYPERTENSIVE MEDICATION |
| 2 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ARTERIAL HYPERTENSION |
| 3 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | BENIGN ESSENTIAL HYPERTENSION |
| 4 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | ESSENTIAL HYPERTENSION |
| 5 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | GRADE 1 HYPERTENSION |
| 6 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HIGH BLOOD PRESSURE |
| 7 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION |
| 8 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION & RIGHT EAR TINNITIS |
| 9 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSION, WORSENING OF |
| 10 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | HYPERTENSIVE CRISIS |

| | Medication Class | Indication |
|---|---|---|
| 11 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | PRESTUDY HYPERTENSION |
| 12 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | STAGE I HYPERTENSION |
| 13 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | UNCONTROLLED HIGH BLOOD PRESSURE |
| 14 | ANTIHYPERTENSIVES | HYPERTENSION |
| 15 | ANTITHROMBOTIC AGENTS | TO THIN THE BLOOD TO TREAT THE INDICATION OF HIGH BLOOD PRESSURE |
| 16 | BETA BLOCKING AGENTS | ARTERIAL HYPERTENSION |
| 17 | BETA BLOCKING AGENTS | BENIGN HYPERTENSION |
| 18 | BETA BLOCKING AGENTS | BITEMPORAL HEADACHE;<br>PRESTUDY HYPERTENSION |
| 19 | BETA BLOCKING AGENTS | ELEVATED BLOOD PRESSURE |
| 20 | BETA BLOCKING AGENTS | HIGH BLOOD PRESSURE |
| 21 | BETA BLOCKING AGENTS | HYPERTENSION |
| 22 | BETA BLOCKING AGENTS | HYPERTENTSION/HEART PALPATATIONS |
| 23 | BETA BLOCKING AGENTS | WORSENING HYPERTENSION |
| 24 | CALCIUM CHANNEL BLOCKERS | ANTI-HYPERTENSIVE MEDICATION |
| 25 | CALCIUM CHANNEL BLOCKERS | ANTIHYPERTENSIVE MED |
| 26 | CALCIUM CHANNEL BLOCKERS | ESSENTENTIAL HYPERTENSION |
| 27 | CALCIUM CHANNEL BLOCKERS | ESSENTILA HYPERTENSION |
| 28 | CALCIUM CHANNEL BLOCKERS | HIGH BLOOD PRESSURE |
| 29 | CALCIUM CHANNEL BLOCKERS | HYPERTENSION |
| 30 | CALCIUM CHANNEL BLOCKERS | PRESTUDY HYPERTENSION |
| 31 | DIURETICS | ARTERIAL HYPERTENSION |
| 32 | DIURETICS | ELEVATED BLOOD PRESSURE |
| 33 | DIURETICS | HIGH BLOOD PRESSURE |
| 34 | DIURETICS | HYPERTENSION |
| 34 | DIURETICS | HYPERTENSION AND EDEMA |
| 36 | DIURETICS | PRESTUDY HYPERTENSION |
| 37 | PERIPHERAL VASODILATORS | HYPERTENSION |

| | Medication Class | Indication |
|---|---|---|
| | Diak | petes |
| 1 | ANALGESICS | DIABETES MELLITUS |
| 2 | ANALGESICS | DIABETIC NEUROPATHY |
| 3 | BLOOD SUBSTITUTES AND PERFUSION SOLUTIONS | DIABETES TYPE II |
| 4 | DRUGS USED IN DIABETES | ADULT ONSET DIABETES MELLITUS |
| 5 | DRUGS USED IN DIABETES | ADULT ONSET DIABETES MELLITUS (TYPE 2) |
| 6 | DRUGS USED IN DIABETES | ADULT ONSET DIABETES MELLITUS TYPE 2 |
| 7 | DRUGS USED IN DIABETES | CONTROL SUGAR |
| 8 | DRUGS USED IN DIABETES | DIABETES |
| 9 | DRUGS USED IN DIABETES | DIABETES (AODM) |
| 10 | DRUGS USED IN DIABETES | DIABETES (HIPERGLICEMIA) |
| 11 | DRUGS USED IN DIABETES | DIABETES II |
| 12 | DRUGS USED IN DIABETES | DIABETES MELLITIS TYPE II |
| 13 | DRUGS USED IN DIABETES | DIABETES MELLITUS |
| 14 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II |
| 15 | DRUGS USED IN DIABETES | DIABETES MELLITUS (ADULT ONSET/TYPE 2) |
| 16 | DRUGS USED IN DIABETES | DIABETES MELLITUS 2 |
| 17 | DRUGS USED IN DIABETES | DIABETES MELLITUS BY HYSTORY |
| 18 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE I WITH<br>HYPERLIPIDEMIA |
| 19 | DRUGS USED IN DIABETES | DIABETES MELLITUS II |
| 20 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE 2 |
| 21 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE II |
| 22 | DRUGS USED IN DIABETES | DIABETES MELLITUS, TYPE II |
| 23 | DRUGS USED IN DIABETES | DIABETES MILLITUS |
| 24 | DRUGS USED IN DIABETES | DIABETES TYPE 1 |
| 25 | DRUGS USED IN DIABETES | DIABETES TYPE 2 |
| 26 | DRUGS USED IN DIABETES | DIABETES TYPE 2 DINOVO |
| 27 | DRUGS USED IN DIABETES | DIABETES TYPE II |
| 28 | DRUGS USED IN DIABETES | DIABETIS |
| 29 | DRUGS USED IN DIABETES | DIABETTES MELLITUS |
| 30 | DRUGS USED IN DIABETES | DM |
| 31 | DRUGS USED IN DIABETES | DM2 |
| 32 | DRUGS USED IN DIABETES | HYPERGLYCEMIA |
| 33 | DRUGS USED IN DIABETES | NONINSULIN-DEPENDENT DIABETES MELLITUS |
| 34 | DRUGS USED IN DIABETES | PRESTUDY DIABETES MELLITUS |
| 34 | DRUGS USED IN DIABETES | TYPE 2 DIABETES |
| 36 | DRUGS USED IN DIABETES | TYPE 2 DIABETES MELLITUS |
| 37 | DRUGS USED IN DIABETES | TYPE II DIABETES |
| 38 | DRUGS USED IN DIABETES | WORSENING OF DIABETES |

| | Medication Class | Indication |
|---|---|---|
| | Cardiovascular Disease | |
| 1 | AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM | NON-ST SEGMENT ELEVATION MYOCARDIAL INFARCTION |
| 2 | ALL OTHER THERAPEUTIC PRODUCTS | WORSENING OF CORONARY ARTERY DISEASE |
| 3 | ANALGESICS | CORONARY ARTERY DISEASE |
| 4 | ANALGESICS | INTERMITTENT CLAUDICATION OF THE LOWER EXTREMITIES |
| 5 | ANALGESICS | ISCHEMIC LEFT TOE |
| 6 | ANALGESICS | ST ELEVATION MYOCARDIAL INFARCTION |
| 7 | ANALGESICS | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 8 | ANALGESICS | STROKE RELATED PAIN |
| 9 | ANALGESICS | STROKE RELATED PAIN (POST-OP) |
| 10 | ANALGESICS | WORSENING OF CORONARY ARTERY DISEASE |
| 11 | ANESTHETICS | ST ELEVATION MYOCARDIAL INFARCTION |
| 12 | ANESTHETICS | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 13 | ANTIANEMIC PREPARATIONS | WORSENING OF CORONARY ARTERY DISEASE |
| 14 | ANTIBACTERIALS FOR SYSTEMIC USE | ST ELEVATION MYOCARDIAL INFARCTION |
| 15 | ANTIBACTERIALS FOR SYSTEMIC USE | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 16 | ANTIEMETICS AND ANTINAUSEANTS | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 17 | ANTIEPILEPTICS | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 18 | ANTIHYPERTENSIVES | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 19 | ANTIHYPERTENSIVES | WORSENING OF CORONARY ARTERY DISEASE |
| 20 | ANTIINFLAMMATORY AND ANTIRHEUMATIC PRODUCTS | STROKE RELATED PAIN |
| 21 | ANTITHROMBOTIC AGENTS | CARDIOVASCULAR ACCIDENT PROPHYLAXIS |
| 22 | ANTITHROMBOTIC AGENTS | CARDIOVASCULAR DISEASE PROPHYLAXIS |
| 23 | ANTITHROMBOTIC AGENTS | CARDIOVASCULAR EVENT PROPHYLAXIS |
| 24 | ANTITHROMBOTIC AGENTS | CARDIOVASCULAR PROPHYLAXIS |
| 25 | ANTITHROMBOTIC AGENTS | CARDIOVASCULRAL PROPHYLAXIS |
| 26 | ANTITHROMBOTIC AGENTS | CORONARY ARTERY DISEASE |
| 27 | ANTITHROMBOTIC AGENTS | CORONARY DISEASE |
| 28 | ANTITHROMBOTIC AGENTS | CORONARY STENTS |
| 29 | ANTITHROMBOTIC AGENTS | HISTORY OF STROKE |
| 30 | ANTITHROMBOTIC AGENTS | ISCHEMIC EVENTS PREVENTION |
| 31 | ANTITHROMBOTIC AGENTS | LEFT VENTRICULAR ISCHEMIA ANTERIOIR |
| 32 | ANTITHROMBOTIC AGENTS | MILD CORONARY ATHEROSCLEROSIS |

| | Medication Class | Indication |
|---|---|---|
| 33 | ANTITHROMBOTIC AGENTS | NON-ST SEGMENT ELEVATION MYOCARDIAL INFARCTION |
| 34 | ANTITHROMBOTIC AGENTS | POST CORONARY ARTERY BYPASS GRAFT |
| 34 | ANTITHROMBOTIC AGENTS | PREVENT CARDIOVASCULAR EVENT |
| 36 | ANTITHROMBOTIC AGENTS | STROKE (BLOOD CLOT PROPHYLAXIS) |
| 37 | ANTITHROMBOTIC AGENTS | STROKE (PROPHYLAXIS) |
| 38 | ANTITHROMBOTIC AGENTS | STROKE PREVENTION |
| 39 | ANTITHROMBOTIC AGENTS | STROKE PROHYLAXIS |
| 40 | ANTITHROMBOTIC AGENTS | TO PREVENT HEART ATTACK/STROKE |
| 41 | ANTITHROMBOTIC AGENTS | VASOSPASTIC ANGINA |
| 42 | ANTITHROMBOTIC AGENTS | WORSENING OF CORONARY ARTERY DISEASE |
| 43 | BETA BLOCKING AGENTS | CARDIOVASCULAR PROTECTION POST INFERIOR WALL MYOCARDIAL INFARCTION |
| 44 | BETA BLOCKING AGENTS | CORONARY ARTERY DISEASE |
| 45 | BETA BLOCKING AGENTS | CORONARY DISEASE |
| 46 | BETA BLOCKING AGENTS | LONG TERM MANAGEMENT OF ANGINA |
| 47 | BETA BLOCKING AGENTS | NON-ST SEGMENT ELEVATION MYOCARDIAL INFARCTION |
| 48 | BETA BLOCKING AGENTS | ST ELEVATION MYOCARDIAL INFARCTION |
| 49 | BLOOD SUBSTITUTES AND PERFUSION SOLUTIONS | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 50 | BLOOD SUBSTITUTES AND PERFUSION SOLUTIONS | WORSENING OF CORONARY ARTERY DISEASE |
| 51 | CALCIUM CHANNEL BLOCKERS | ST ELEVATION MYOCARDIAL INFARCTION |
| 52 | CALCIUM CHANNEL BLOCKERS | VASOSPASTIC ANGINA |
| 53 | CARDIAC THERAPY | CORONARY ARTERY DISEASE |
| 54 | CARDIAC THERAPY | NON-ST SEGMENT ELEVATION MYOCARDIAL INFARCTION |
| 55 | CARDIAC THERAPY | WORSENING OF CORONARY ARTERY DISEASE |
| 56 | DIURETICS | ST ELEVATION MYOCARDIAL INFARCTION |
| 57 | DRUGS FOR ACID RELATED DISORDERS | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 58 | DRUGS FOR FUNCTIONAL GASTROINTESTINAL DISORDERS | ST ELEVATION MYOCARDIAL INFARCTION (STEMI) |
| 59 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE |
| 60 | LIPID MODIFYING AGENTS | LEFT VENTRICULAR ISCHEMIA |
| 61 | LIPID MODIFYING AGENTS | STROKE PREVENTION |
| 62 | MINERAL SUPPLEMENTS | WORSENING OF CORONARY ARTERY DISEASE |
| 63 | PERIPHERAL VASODILATORS | CORONARY ARTERY DISEASE |
| 64 | PSYCHOLEPTICS | ST ELEVATION MYOCARDIAL INFARCTION |
| 65 | PSYCHOLEPTICS | WORSENING OF CORONARY ARTERY DISEASE |
| 66 | STOMATOLOGICAL PREPARATIONS | ANGINA |
| 67 | VITAMINS | WORSENING OF CORONARY ARTERY DISEASE |

| | Medication Class | Indication | | | |
|---|---|---|--|--|--|
| | Hyperlipidemia | | | | |
| 1 | ANTITHROMBOTIC AGENTS | HYPERLIPIDEMIA | | | |
| 2 | DRUGS USED IN DIABETES | DIABETES MELLITUS TYPE I WITH<br>HYPERLIPIDEMIA | | | |
| 3 | GENERAL NUTRIENTS | HYPERTRIGLYCERIDEMIA | | | |
| 4 | LIPID MODIFYING AGENTS | ACUTE MIOCARDIAL INFARCTION | | | |
| 5 | LIPID MODIFYING AGENTS | ANAL FISSURE | | | |
| 6 | LIPID MODIFYING AGENTS | ANTIHYPERLIPIDEMIA PROPHYLAXIS | | | |
| 7 | LIPID MODIFYING AGENTS | CHOLESTEROLEMIA | | | |
| 8 | LIPID MODIFYING AGENTS | CORONARY ARTERY DISEASE | | | |
| 9 | LIPID MODIFYING AGENTS | DIABETES MELLITUS TYPE I WITH<br>HYPERLIPIDEMIA | | | |
| 10 | LIPID MODIFYING AGENTS | DIETARY SUPPLEMENT | | | |
| 11 | LIPID MODIFYING AGENTS | DYSLIPIDEMA | | | |
| 12 | LIPID MODIFYING AGENTS | DYSLIPIDEMIA | | | |
| 13 | LIPID MODIFYING AGENTS | DYSLIPIDEMIE | | | |
| 14 | LIPID MODIFYING AGENTS | FUNCTIONAL DIARRHEA | | | |
| 15 | LIPID MODIFYING AGENTS | GENERAL HEALTH | | | |
| 16 | LIPID MODIFYING AGENTS | GENERAL NUTRITION | | | |
| 17 | LIPID MODIFYING AGENTS | HEALTH MAINTENANCE | | | |
| 18 | LIPID MODIFYING AGENTS | HEALTH SUPPLEMENT | | | |
| 19 | LIPID MODIFYING AGENTS | HEALTH SUPPLEMENTS | | | |
| 20 | LIPID MODIFYING AGENTS | HIGH BLOOD PRESSURE | | | |
| 21 | LIPID MODIFYING AGENTS | HIGH CHOLESTEROL | | | |
| 22 | LIPID MODIFYING AGENTS | HISTORY OF DYSLIPIDEMIA | | | |
| 23 | LIPID MODIFYING AGENTS | HISTORY OF MIX HYPERLIPIDEMIA | | | |
| 24 | LIPID MODIFYING AGENTS | HUMAN PAPILLOMAVIRUS (RECTAL) | | | |
| 25 | LIPID MODIFYING AGENTS | HYPELIPIDEMIA | | | |
| 26 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLAEMIA | | | |
| 27 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMAIL | | | |
| 28 | LIPID MODIFYING AGENTS | HYPERCHOLESTEROLEMIA | | | |
| 29 | LIPID MODIFYING AGENTS | HYPERGLYCERIDEMIA | | | |
| 30 | LIPID MODIFYING AGENTS | HYPERLIDPDEMA | | | |
| 31 | LIPID MODIFYING AGENTS | HYPERLIPDEMIA | | | |
| 32 | LIPID MODIFYING AGENTS | HYPERLIPEDEMIA | | | |
| 33 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA | | | |
| 34 | LIPID MODIFYING AGENTS | HYPERLIPIDEMIA WORSENED | | | |
| 34 | LIPID MODIFYING AGENTS | HYPERLIPIEMIA | | | |
| 36 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERICEMIA | | | |
| 37 | LIPID MODIFYING AGENTS | HYPERTRIGLYCERIDEMIA | | | |
| | Medication Class | Indication |
|---|---|---|
| 38 | LIPID MODIFYING AGENTS | INCREASED LIPIDS |
| 39 | LIPID MODIFYING AGENTS | MIXED HYPERLIPIDEMIA |
| 40 | LIPID MODIFYING AGENTS | NUTITIONAL SUPPLEMENT |
| 41 | LIPID MODIFYING AGENTS | NUTRITIONAL SUPPLEMENT |
| 42 | LIPID MODIFYING AGENTS | NUTRITIONAL SUPPLEMENTS |
| 43 | LIPID MODIFYING AGENTS | PREVENTATIVE |
| 44 | LIPID MODIFYING AGENTS | STROKE PREVENTION |
| 45 | LIPID MODIFYING AGENTS | SUPLLEMENT |
| 46 | LIPID MODIFYING AGENTS | SUPPLEMENT |
| 47 | LIPID MODIFYING AGENTS | SUPPLEMENTATION |
| 48 | LIPID MODIFYING AGENTS | TACHYARRHYTHMIA |
| 49 | LIPID MODIFYING AGENTS | WELLNESS |
| 50 | LIPID MODIFYING AGENTS | WORSENING HYPERCHOLESTEROLEMIA |
| 51 | UNSPECIFIED HERBAL AND TRADITIONAL MEDICINE | HYPERCHOLESTEROLEMIA |

## **Appendix 7. Programming Specification**

#### **General Conventions**

- 1) The standard mock tables (http://gnet/biometrics/stat/doc/Standard%20TFL\_Final%20GNET%202009%2005%2015.doc) are default outputs developed based on standard CRF and standard SAP template. Changes to the CRFs or SAP may warrant changes to these outputs.
- 2) Italicized text in the mocks indicates that the entry is either optional or can be replaced by a more suitable term depending on the content.
- 3) Whenever possible, do not reference footnote by symbol within the body of the table and table title unless it greatly improves the clarity.
- 4) Titles should not exceed 128 characters (including the word "table," the table number, punctuation, and spaces). If a title must exceed 128 characters, key descriptive information should be presented in the first 128 characters.
- 5) For completeness, please always include all the possible categories on standard CRF, including those with zero counts.
- 6) Treatment groups will be ordered as Gilead product in the first and then the rest of active control groups in alphabetical order, and placebo in the last column. Within each treatment, dose level will be in ascending order. Separate column for total or subtotal are allowed if space permits depending on study design, eg, a subtotal column could combine dose levels within the same treatment.
- 7) The ordering of these mock tables is the default ordering in the TFLs, ie, enrollment, disposition, demographic, baseline data, efficacy, drug exposure, and safety.
- 8) Number TFLs consecutively and do not use decimal numbering for unique items.
- 9) A maximum of three titles and seven footnotes is allowed. Additional lines document the date of date extraction, source of SAS program, output files, and date-time of outputs generated.
- 10) The precision in reporting numerical values should be as follows:
  - a) Raw measurements will be reported the same as the data captured electronically or on the CRFs.
  - b) Standard deviation and stand error will be reported to one more significant decimal place than the raw measurement.
  - c) Mean, median, minimum, Q1, Q3, maximum, 95% CIs will be reported to the same number of decimal places of the raw measurements.
  - d) Exceptions may be considered; for example if more than 4 significant digits are provided for the measurement.

- 11) The number of decimal places in reporting p-values should be as follows:
  - a) values less than  $0.001 \rightarrow <0.001$
  - b) values 0.001 to less than  $0.10 \rightarrow$  round to 3 decimal places
  - c) values 0.10 and greater  $\rightarrow$  round to 2 decimal places
- 12) For lab summaries, tests will be grouped as Chemistry, Hematology, and Metabolic Assessments. Disease related biomarkers, eg, bone biomarkers, will be grouped separately. Summaries will be sorted alphabetically by test within group.
- 13) Study day: if visit date ≥ first dose date, study day = visit date first dose date +1. If visit date < first dose date, study day = visit date first dose date.

#### Other Definitions

- 1) AGE calculated as follows:
  - a) AGE (years) is calculated from the number of days between the date of birth (DOB) and Day 1 (first dose date),
  - b) Use the SAS INTCK function to determine the number of "1st-of-month days" (eg, January 1st, February 1st, March 1st) between DOB and Day 1 (inclusive),
  - c) Divide the result in (b) by 12,
  - d) AGE = the integer of the result in (c),
  - e) If the DOB and Day 1 have the month in common and the birthday is later in the month than the date of Study Day 1, subtract one from the AGE result above.

For subjects randomized and never dosed with study drug, age will be calculated from the date of randomization.

- 2) All screened subjects refer to all subjects who are screened (ie, with nonmissing screening date) and have a screening number. For summarization, same subject is counted only once. DOB and other demographic information such as sex, race, and ethnicity, country and initials will be used for identifying unique screened subjects.
- 3) Screen failure subjects are the subjects who are screened and answered "No" for any inclusion criteria or "Yes" for any exclusion criteria regardless of which version of protocol the subject was consent to.
- 4) Subjects in the randomized analysis set are defined as subjects randomized into the study. IXRSRAND is the source to determine whether the subject is randomized (ie, subject with nonmissing RGMNDTN in the IXRSRAND dataset) and confirmed by the eCRF ENROLL dataset (ie, ENROLLYN = "Yes" in ENROLL dataset).

- 5) In disposition table, the reasons for premature discontinuation are displayed in the order as they appear on the eCRF.
- 6) Body mass index (BMI)

Calculated from height in meters (eg, height in cm/100) and weight in kilograms as:

BMI will be calculated only at baseline. Baseline height and weight will be used for the BMI = (weight [kg])/ (height [meters]<sup>2</sup>) calculation (height will be obtained from Vital Signs eCRF at screening visit, weight will be obtained from Vital Signs eCRF at baseline visit, if it's missing, weight at screening visit from Vital Signs eCRF will be used).

- 7) Please note, "Not Permitted" or missing categories will be excluded for p value generation for categorical data analysis (eg, CMH test or Fisher exact test).
- 8) HIV Tagman Calculations

If a HIV-1 RNA test value is reported as "< 20 cp/mL HIV-1 RNA Detected" or "No HIV-1 RNA detected", a numeric value of 19 will be used for summary purpose.

- 9) For safety ECGs at postbaseline visits, the most conservative (worst) value within the window will be selected, eg, abnormal will be selected over normal for safety ECG or clinically significant abnormal will be selected over not clinically significant abnormal if there are multiple abnormal findings.
- 10) SAS codes for treatment comparison for demographics and baseline characteristics tables.
  - a) CMH test for nominal variable (Y):

```
proc freq order=data;
   tables treat * Y /cmh /*general association test*/
run;
```

b) CMH test for ordinal variable (Y):

```
proc freq order=data;
   tables treat * Y / cmh2 ; /*row mean score test*/
run;
```

c) Wilcoxon rank sum test for continuous variable (Y):

```
proc npar1way wilcoxon data=xxxx;
   class treat;
   var Y;
run;
```

11) SAS codes for treatment comparison using Fisher's exact test

```
proc freq order=adsl;
   tables trtgrp * Y /fisher riskdiff;
run;
```

## 12) Last Dose Date and Last Study Date

- a) Last Dose Date (ie, TRTEDTC or TRTEDT in ADSL)
  - i) For subjects on E/C/F/TAF or delayed switch to E/C/F/TAF:
    - For subjects with a partial last dosing date (ie, month and year of last dose are known), use the max (the dispensing dates of study drug bottles, study drug start dates and end dates, imputed last dose date [day imputed as 15]) as the final imputed last dose date. (However if dispensing date's month is after last dose date's month, data query is needed.)
    - If subject died and the death date is complete (ie, not partial date) and before the imputed last dose date, the complete death date should be used as the imputed last dose date.
    - If the date of last dose is missing (eg, only year of last dose is known or completely missing due to lost to follow-up), use the maximum of study drug start dates and end dates, clinic visit dates (i.e., visit dates from vital sign and ECG forms), and laboratory visit dates excluding the 30-day follow-up visit to impute the last dose date.
  - ii) For subjects taking ABC/3TC+3rd Agent:
    - For subjects with a partial last dose date (ie, month and year of last dose are known) or missing last dose date (ie, only year of last dose is known or completely missing due to lost to follow-up):
      - If the subject has an E/C/F/TAF start date and if the month and year of the last dose date are the same as the start date of E/C/F/TAF, then the last dose date will be set to the start date of E/C/F/TAF − 1.
      - If the subject does not have an E/C/F/TAF start date, then use the maximum of clinic visit dates (i.e., visit dates from vital sign and ECG forms), and laboratory visit dates excluding the 30-day follow-up visit to impute the last dose date.
- b) Last Study Date is the maximum of nonmissing study drug start dates and end dates, clinic visit dates (i.e., visit dates from vital sign and ECG forms) and laboratory visit dates, including the 30-day follow-up visit date for subjects who prematurely discontinued study or who completed study according to study completion eCRF. Please note, if study drug start date or end date is partially missing, the imputed date (day imputed as 15) will be used. If subject died and the death date is complete (ie, not partial date) and before the imputed last study date, the complete death date should be used as the imputed last study date.

## 13) Toxicity Grades:

- a) For toxicity grade summary, we will include all postbaseline graded results up to 30 days after last dose of study drug, not just those at summarized visits.
- b) For hematuria grading, if the laboratory reports urine blood using the plus system (+1, +2, etc) and also provides quantitative results on reflex (ie, urine RBC), summarize only the grade of the urine RBC results, but list both grades of urine blood and urine RBC.
- c) For glucose grading, as specified in SAP Section 7.2.2.1, the treatment-emergent flag cannot be determined for nonfasting glucose (including glucose results without a known fasting status). As a result, these records will be excluded from the "Maximum Treatment-emergent Toxicity Grade" summary in the "Treatment-emergent Laboratory Abnormalities" or "Treatment-emergent Grade 3 or 4 Laboratory Abnormalities" summary tables. In addition, fasting glucose and nonfasting glucose will be listed as two separate laboratory tests in the "Laboratory Abnormalities" and "Grade 3 or 4 Laboratory Abnormalities" listings. Only a maximum postbaseline toxicity flag will be displayed and the treatment-emergent flag will not be displayed for nonfasting glucose as the treatment-emergent flag cannot be determined for nonfasting glucose.

## 14) "On-treatment" means the following for each treatment group

- a) For efficacy data (eg, HIV-1 RNA (snapshot algorithm) and CD4) in the SAP:
  - i) For E/C/F/TAF, data collected up to 1 day after the last dose date of study drug
  - ii) For ABC/3TC + 3rd Agent, data collected up to 1 day after the last dose date of ABC/3TC + 3rd Agent
  - iii) For Delayed Switch E/C/F/TAF, data collected from the first dose date of E/C/F/TAF up to 1 day after the last dose date of study drug
- b) For safety data (Proteinuria by Dipstick [Section 7.4.3], UPCR and UACR [Section 7.4.4], RBP to Creatinine Ratio and Beta-2-Microglobulin to Creatinine Ratio [Section 7.4.5]) in the SAP:
  - i) For E/C/F/TAF, data collected up to 1 day after the last dose date of study drug
  - ii) For ABC/3TC + 3rd Agent, data collected up to 1 day after the last dose date of ABC/3TC + 3rd Agent
  - iii) For Delayed Switch E/C/F/TAF, data collected from the first dose date of E/C/F/TAF up to 1 day after the last dose date of study drug

- c) For all other safety data in the SAP:
  - i) For E/C/F/TAF, data collected up to 30 days after the last dose date of study drug
  - ii) For ABC/3TC + 3rd Agent, data collected up to the minimum of (1) the last dose date of ABC/3TC+3rd Agent plus 30 days or (2) the first dose date of E/C/F/TAF
  - iii) For Delayed Switch E/C/F/TAF, data collected from the first dose date of E/C/F/TAF up to 30 days after the last dose date of study drug

#### 15) Efficacy analyses:

a) Exact method for difference in primary endpoint or other efficacy endpoints with proportion of HIV-1 RNA <50 c/mL between treatment group: the code below provides exact CIs (on an unconditional exact method using 2 inverted 1-sided tests) in SAS v9.3 or above:

```
data example;
  input trt01a $ outcome $ count;
  datalines;
Treat-A
             2-Fail
Treat-A
             1-Succ
                         189
Treat-B
Treat-B
             2-Fail
1-Succ
                           4
                            88
run;
proc freq data = example noprint;
  table trt01a*outcome /riskdiff(CL=(exact)) alpha=0.05;
  weight count; exact RISKDIFF(METHOD=SCORE);
  output out=ciexact(keep= RDIF1 XL RDIF1 XU RDIF1) riskdiff;
run;
data final (keep=Estimate LowerCL UpperCL ocharc1);
  set ciexact;
  label Estimate ="Percentage Difference"
        LowerCL = "95% Lower Confidence Limit"
        UpperCL = "95% Upper Confidence Limit";
  Estimate=100* RDIF1;
  LowerCL = 100*XL RDIF1;
  UpperCL = 100*XU RDIF1;
  ocharc1 = right(compress(put(Estimate, 8.1)) || '% (' ||
compress(put(LowerCL,8.1)) || '% to ' || compress(put(UpperCL,8.1)) ||
'%)');
run;
```

b) ANOVA model for continuous efficacy variable (eg, CD4):

The differences in changes from baseline in CD4 cell count between treatment groups and the associated 95% CI will be constructed using ANOVA, including treatment as a fixed effect in the model.

SAS code is as follows:

```
proc glm data=adeff;
   class trtgrp;
   model CD4=trtgrp;
   lsmeans trtgrp /alpha=0.05 cl pdiff;
run;
```

c) Listing for snapshot algorithm outcome:

In addition to flagging the values of HIV-1 RNA < 50 or  $\ge 50$  for snapshot algorithm virologic outcomes, flag the last available HIV-1 RNA value for the following categories:

- i) HIV-1 RNA >= 50 copies/mL Discontinued Study Drug Due to AE or Death and Last Available HIV-1 RNA >= 50 copies/mL
- ii) HIV-1 RNA >= 50 copies/mL Discontinued Study Drug Due to Other reason\* and Last Available HIV-1 RNA >= 50 copies/mL
- iii) No virologic Data Discontinued Study Drug Due to AE or Death and Last Available HIV-1 RNA < 50 copies/mL
- iv) No virologic Data Discontinued Study Drug Due to Other reason\* and Last Available HIV-1 RNA < 50 copies/mL
- Note: \* Other reasons include subjects who discontinued study drug due to investigator's discretion, subject decision, lost to follow-up, noncompliance with study drug, protocol violation, pregnancy, and study terminated by sponsor.
- 16) Treatment-emergent proteinuria analyses with rank analysis of covariance

```
proc rank data=up nplus1 ties=mean out=ranks1;
   var upbase upwk48;
run;

proc reg data=ranks1;
   model upwk48=upbase;
   output out=residual1 r=resid;
run;

proc freq data=residual1;
   tables trtgrp*resid/noprint cmh2;
run;
```

#### 17) TEAE

#### **Events with Missing Onset Day and/or Month**

The event is treatment emergent if the following 3 criteria are met:

- The month and year (or year) of onset date is the same as or after the month and year (or year) of the first dose of study drug, and
- The month and year (or year) of the onset date is the same as or before the month and year (or year) of 30th day after the date of the last dose of study drug, and
- End date is as follows:
  - The (complete) end date is on or after the first dose date, or
  - The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of study drug, or
  - End date is completely missing

## **Events with Completely Missing Onset Date**

An AE with a completely missing onset date is defined as TEAE if end date is as follows:

- The (complete) end date is on or after the first dose date, or
- The month and year (or year) of end date is the same or after the month and year (or year) of the first dose of study drug, or
- End date is completely missing

## **Events in Treatment Arm 2 with Ambiguous Onset Date**

For subjects in Treatment Arm 2, an AE with a partial date that shares the same month and year (or year only if month is missing) with the end date of ABC/3TC + 3rd Agent and the start date of E/C/F/TAF will be considered to be treatment-emergent for E/C/F/TAF

#### **Events Leading to Study Drug Discontinuation in Treatment Arm 2**

For subjects in Treatment Arm 2, an AE that leads to study drug discontinuation will be considered treatment-emergent for the period in which the discontinuation occurs. If the AE starts while subject is on ABC/3TC + 3rd Agent and leads to discontinuation while on E/C/F/TAF, then it will be considered treatment-emergent for both ABC/3TC + 3rd Agent and E/C/F/TAF.

## 18) Urine Protein Correction

a) The calibrator material used in the quantitative assay for the measurement of urine protein (UP) was changed globally in Covance on May 27, 2016. All samples reported prior to May 27, 2016 (ie, *RPTDTM* < 'May 27, 2016') were tested by the calibrator material manufactured by Roche Diagnostics, while the samples reported on or after May 27, 2016 were tested by the calibrator material manufactured by Quantimetrix. Covance had 3 regional lab centers to run the samples. Each regional lab center conducted its own alternate (quantitative) method comparison. These comparisons demonstrate that calibrator materials manufactured by the Roche and Quantimetrix yield comparable results as noted in the table below:

| Regional Lab Center | Accession Numbers <sup>a</sup> | Regular Regression for UP Correction <sup>b</sup> | Correlation<br>Coef. | Bias |
|---|---|---|---|---|
| Indianapolis Auto<br>Chemistry | Start with 65 | Y = 1.028 X - 3.70 | 0.9982 | -2.34 (-4.91%) |
| Geneva Auto Chemistry | Start with 62 or 63 | Y = 0.981 X - 1.44 | 0.9993 | -2.42 (-4.74%) |
| Singapore Auto<br>Chemistry | Start with 64 or 66 | Y = 0.980 X - 1.62 | 0.9996 | -2.73 (-5.08%) |
| BML in China | Start with 67 or 68 | NA | NA | NA |

a Accession numbers specified which regional lab center tested the sample. For example, samples with accession number started with 65 were tested in Indianapolis Auto Chemistry Center.

b X and Y are the UP results using calibrator materials manufactured by Roche Diagnostics and Quantimetrix, respectively.

| b) | In order to combine the UP results obtained from the 2 different assay methods for |
|---|---|
| | summary/comparison, we will convert the UP results analyzed using the calibrator from |
| | Roche (ie, results reported prior to May 27, 2016) to Quantimetrix results by using the |
| | regression equation listed in the above table. |

| Original UP based on Reported Date | Original UP<br>Categories | Accession<br>Number | AVALC of Corrected UP<br>('UP' stands for Original UP) |
|---|---|---|---|
| UP reported on/after<br>May 27, 2016 | _ALL_ | _ALL_ | AVALC of UP |
| | UP < 4.0 | _ALL_ | '< 4.0' |
| LID noncentral historia | | Start with 65 | 1.028 × LIP = 3.70 · if 1.028 × LIP = 3.70 > 4.0 |
| UP reported before May 27, 2016 | $\mathrm{UP} \geq 4.0$ | Start with 62 or 63 | $0.981 \times UP - 1.44$ ; if $0.981 \times UP - 1.44 \ge 4.0$ '< $4.0$ '; if $0.981 \times UP - 1.44 < 4.0$ |
| | | Start with 64 or 66 | $0.980 \times UP - 1.62$ ; if $0.980 \times UP - 1.62 \ge 4.0$<br>'< $4.0$ '; if $0.980 \times UP - 1.62 < 4.0$ |

c) The corrected UP results will be used for the following analysis and referred as "UP" in following text. If AVALC of the corrected UP is "< 4.0", the AVAL of the corrected UP will be imputed as 3.9 mg/dL.

- 19) Unit conversion for some renal biomarkers derived from related tests with conventional units
  - Urine RPB ( $\mu$ g/L) to creatinine (mg/dL) ratio: 1 ( $\mu$ g/L) / (mg/dL) = 100 ×  $\mu$ g/g
  - Urine Beta-2-microglobulin (mg/L) to creatinine (mg/dL) ratio:  $1 \text{ (mg/L)} / \text{ (mg/dL)} = 10^5 \text{ µg/g}$
  - Urine Protein (mg/dL) to creatinine (mg/dL) ratio:  $1 \text{ (mg/dL)} / \text{ (mg/dL)} = 1000 \times \text{mg/g}$
  - Urine Albumin (mg/dL) to creatinine (mg/dL) ratio:  $1 \text{ (mg/dL)} / \text{ (mg/dL)} = 1000 \times \text{mg/g}$

## 20) Calculation of ratios

To calculate laboratory ratios (eg, urine RPB to creatinine ratio), lab value of each test in the ratio needs to be from the same accession number; if any test value used for the ratio calculation from the same accession number is missing, the ratio is not calculable (ie, missing). For urine creatinine, a value of "< 1" is handled as a missing value in the calculation of related ratios. For urine protein, a value of "< 4.0" is handled as a missing value in the calculation of UPCR.

- 21) Combined category of UP and UPCR
  - a) First merge UP and UPCR based on the subject identifier and accession number.
  - b) At each visit, based on UP to select which pair of records should be used for the analysis. That is, once a UP record is selected for that visit, the UPCR with the same accession number (if calculated) will be selected. Please note, UPCR is missing when UP < 4.0 mg/dL.
  - c) Subject will be classified as "UPCR ≤ 200 mg/g" if UP < 4.0 mg/dL or UPCR ≤ 200 mg/g; Subject will be classified as "UPCR > 200 mg/g" if UPCR > 200 mg/g; Otherwise, subject will be classified as "Missing".

#### 22) Prior ARV

Non-study drug ARVs collected in prior ARV form with start date and stop date completely missing are considered "not concomitant".

- 23) Age for laboratory test reference range will be based on the age at the sample collection date.
- 24) For figures, if at a visit where n (sample size) for any treatment group <= 5, data for that treatment group will not be displayed at the visit in figure, but all data will be included in the corresponding table summary.
- 25) For PRO data, data up to 30 days after the last dose date for subjects who permanently discontinued study drug will be summarized.

26) For PRO data, unless otherwise stated, multiple responses and out of range responses will be set to missing and missing responses will not be imputed.

Out of range value is determined based on the following table for within-range response values:

SF-36v2 Health Survey:

| | Response | |
|---|---|---|
| Question | Min | Max |
| 1, 2, 4a to 4d, 5a to 5c, 6, 8, 9a to 9i, 10, 11a to 11d | 1 | 5 |
| 3a to 3j | 1 | 3 |
| 7 | 1 | 6 |

## VAS adherence questionnaire:

| | Resp | Response |
|-----------|------|----------|
| Questions | Min | Max |
| 1 | 0 | 100 |
| 2 | 0 | 30 |
| 3 | 0 | 4 |

27) SAS codes for ANOVA model for analyzing treatment satisfaction questionnaire (HIVTSQc) with baseline status questionnaire (HIVTSQs) as a covariate

```
proc glm data=adeff;
   class trtgrp;
   model hivtsqc = hivtsqs trtgrp hivtsqs* trtgrp;
   /* delete int. term if int. term is not significant ie p > 0.05*/
   lsmeans trtgrp /alpha=0.05 cl pdiff;
run;
```

#### 28) Computing EQ-5D index values with SAS using the UK TTO value set

The variables for the 5 dimensions of the EQ-5D descriptive system should be named 'mobility', 'selfcare', 'activity', 'pain', and 'anxiety'. The variable 'UK\_TTO' contains the values of the EQ-5D index.

You can copy and paste the syntax below directly into the SAS syntax window.

```
***************
* SAS syntax code for the computation of index *
* values with the UK MVH-A1 TTO value set *
*******************
data Eurogol. Uk data;
set Eurogol.EQ5D states;
UK TTO = 1;
if (mobility = 2) then UK TTO = UK TTO - 0.069;
if (mobility = 3) then UK TTO = UK TTO - 0.314;
if (selfcare = 2) then UK TTO = UK TTO - 0.104;
if (selfcare = 3) then UK TTO = UK TTO - 0.214;
if (activity = 2) then UK TTO = UK TTO - 0.036;
if (activity = 3) then UK TTO = UK TTO - 0.094;
if (pain = 2) then UK TTO = UK TTO - 0.123;
if (pain = 3) then UK TTO = UK TTO - 0.386;
if (anxiety = 2) then UK TTO = UK TTO - 0.071;
if (anxiety = 3) then UK TTO = UK TTO - 0.236;
if (mobility ne 1) or (activity ne 1) or (selfcare ne 1) or (pain ne 1) or
(anxiety ne 1) then UK TTO = UK TTO - 0.081;
if (mobility = 3) or (selfcare = 3) or (activity = 3) or (pain = 3) or
(anxiety = 3) then UK TTO = UK TTO - 0.269;
if (mobility = .) or (selfcare = .) or (activity = .) or (pain = .) or
(anxiety = .) then UK TTO = .;
output;
run;
```

## 29) Defining ARV Regimen at Baseline

All subjects are expected to enter the study on ABC/3TC + 3rd Agent, where the 3rd Agent can consist of a drug (possibly with a booster) that is not in the nucleos(t)ide reverse transcriptase inhibitor (NRTI) class. (Note: ABC/3TC consists of 2 NRTI drugs.)

Using the ARV rawdataset, include all prior and/or current ARVs (ARV.INGRED where ARV.CMSCAT ='Prior ARV" or "Current ARV"), taken on or up to 2 days prior to first dose date as defined in Section 3.8.1.

When determining the baseline ARV regimen, please use the following rules:

• The baseline ARV will be recorded as 3rd Agent + ABC/3TC (note the reversed order, as this is due to clinical trials evaluating novel 3rd agents). When ordering the 3rd Agent medications, use the following order to assign priority:

| INGRED | Priority | INGRED | Priority |
|-------------|----------|---------|----------|
| DTG_ABC_3TC | 1 | EFV | 4.1 |
| ATV_COBI | 2.1 | ETR | 4.2 |
| DRV_COBI | 2.2 | NVP | 4.3 |
| LPV_RTV | 2.3 | RPV | 4.4 |
| ATV | 2.4 | ABC_3TC | 5.1 |
| DRV | 2.5 | ABC | 5.2 |
| COBI | 2.6 | 3TC | 5.3 |
| RTV | 2.7 | | |
| DTG | 3.1 | | |
| RAL | 3.2 | | |

- For all ingredients, replace "\_" with "/"
- Make the following replacements to the ingredients:
  - Replace "DTG/ABC/3TC" with "ABC/DTG/3TC"
  - Replace "ATV/COBI" with "ATV/co"
  - Replace "DRV/COBI" with "DRV/co"
  - Replace "LPV/RTV" with "LPV/r"
- Once the ingredients have been updated and assigned an appropriate priority, transpose the ingredients (by subject) and concatenate each column with a "+" following the priority specified above

To illustrate these rules, suppose a subject is on ATV, RTV, and ABC\_3TC. This would translate into "ATV+RTV+ABC/3TC". If, instead, the subject was on LPV\_RTV and ABC\_3TC, their regimen would be presented as "LPV/r+ABC/3TC".

Note: The following data issues should be queried:

- If the subject does not have ABC/3TC (or ABC+3TC) in their baseline regimen
- If a subject does not have a 3rd agent (eg, is only identified as being on ABC/3TC)
- If a subject is on RTV but is not also on ATV or DRV
- If an ARV medication that starts within 30 days of the first dose date (this represents a change in the baseline regimen and would represent an eligibility criteria violation)

### 30) Smoking status at baseline

Smoking status at baseline (ie, never smoker, former smoker, and current smoker) will be summarized as part of the baseline disease characteristics. How to classify a subject as never, former, or current smoker at baseline is specified as follows:

- a) First, select only records with *Type of Substance Use* = "Cigarettes" or "Cigars". Records with *Type of Substance Use* = "Other" (including chew tobacco, e-cigarettes, etc) will not be considered as smoking.
- b) Second, for each selected substance use record, flag whether it is "Prior", "Present", or "Post" relative to the first dose date according to the Algorithm below.
- c) Finally, (1) the subject will be flagged as "Never smoker", if the subject has no record with *Type of Substance Use* = "Cigarettes" or "Cigars" or all selected records have a flag of "Post"; (2) the subject will be flagged as a "Former" smoker, if any selected records has a flag of "Prior" and no record of "Present"; (3) Otherwise, the subject will be flagged as a "Current" smoker, if any selected records has a flag of "Present".

| | Selected Substance Use Records | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Prior | No | No | Yes | Yes | Yes | No | No | Yes |
| Present | No | No | No | No | Yes | Yes | Yes | Yes |
| Post | No | Yes | No | Yes | No | No | Yes | Yes |
| Smoking Status | Never | Never | Former | Former | Current | Current | Current | Current |

# Algorithm to flag whether a selected record is "Prior", "Present", or "Post" relative to the first dose date:

- 1) the start and stop dates of the selected record are not completely missing (ie, at least year is known) or the start date is not missing and record is ongoing. The completed start or stop dates will be used to compare with the first dose date whenever possible. Otherwise, the month and year (or year alone if month is not recorded) of the start or stop dates will be used to compare with the first dose date when the start or stop date of the selected record is incomplete.
  - a) The record is flagged as "Prior", if the stop date is before (<) the first dose date;
  - b) The record is flagged as "Present", if the start date is on or before (≤) the first dose date and the stop date is on or after (≥) the first dose date, or the selected record is marked as ongoing and the start date is on or before (≤) the first dose date;
  - c) The record is flagged as "Post", if the start date is after the first dose date;
- 2) the start date of the selected record is completely missing. We assume that the start date is before the first dose date, the stop date (or the month and/or year of the stop date, if stop date is incomplete) will be used to determine whether the selected record is "Prior" or "Present" as follows.
  - a) The record is flagged as "Prior", if the stop date is before (<) the first dose date or the stop date is completed missing and the record is not marked as ongoing.
  - b) The record is flagged as "Present", if the stop date is on or after (≥) the first dose date or the selected record is marked as ongoing.
- 3) the start date of the selected record is before (<) the first dose date, but the stop date is completely missing and the record is not marked as ongoing. We assume that the end date is before the first dose date, the record is flagged as "Prior".
- 4) the start date of the selected record is on or after the first dose date, but the stop date is completely missing and the record is not marked as ongoing. This is a data issue, should be queried first. However, this record is flagged as "Present" if the start date is on the first dose; this record is flagged as "Post" if the start date is after the first dose.